CLINICAL TRIAL: NCT04143217
Title: An Open-Label Extension Study to Evaluate the Long-Term Safety and Efficacy of SPN-812 (Viloxazine Extended-release Capsule) in Adults With Attention-Deficit/Hyperactivity Disorder
Brief Title: Open-label Long-Term Safety and Efficacy of SPN-812 (Viloxazine Extended-release Capsule) in Adults With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 812P311
Record Dates: First submitted 2019-10-24; First posted 2019-10-29 (Actual); Results first posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label Treatment (Experimental): SPN-812 Open-Label Treatment 200mg to 600mg SPN-812 once daily for up to 156 weeks
  Interventions: Drug: SPN-812

INTERVENTIONS:
Drug: SPN-812 — SPN-812 200 to 600 mg/day
  Other Names: viloxazine extended-release capsules (Qelbree)

SUMMARY:
Open label, flexible dose, long-term multicenter study of safety and efficacy of SPN-812 in adult ADHD patients

DETAILED DESCRIPTION:
This is a multicenter, open-label extension study aimed to assess long-term safety and efficacy of SPN-812 when administered alone or in conjunction with an Food and Drug Administration (FDA)-approved Attention-Deficit Hyperactivity Disorder (ADHD) medication in the treatment of ADHD in adult subjects who completed a blinded study of SPN-812 (812P306). Subjects initiate SPN-812 dosing at 200 mg/day once daily (QD) during first 2 weeks. At or after Visit 2 (Week 2), per the Investigator's discretion and based on Investigator's assessment of subject's clinical response and tolerability, the dose of SPN-812 can be titrated up or tapered down in increments of 50 mg/day, 100 mg/day, 150 mg/day, or 200 mg/day per week to a target dose within the ranges between 200 and 600 mg/day. Additionally, after 12 weeks of dosing (after Visit 4), at the discretion of the Investigator and based on subject's clinical response, the optimized dose of SPN-812 may be supplemented with an adjunctive FDA-approved stimulant treatment. Total treatment duration per subject from Visit 1 to Visit 22 (end of study) is approximately 3 years (156 weeks ± 1 week) or until SPN-812 becomes commercially available.

ELIGIBILITY:
*Please note, Inclusion/Exclusion Criterion "A" applies to subjects who completed Study 812P306 and enrolled in Study 812P311 on either the same day or up to 7 days after the end of Study 812P306. Inclusion/Exclusion Criterion "B" applies to subjects who completed Study 812P306, but enrolled in study 812P311 greater than 7 days after the end of study 812P306*

Inclusion Criteria "A"

1. Is a male or female who completed Study 812P306 and opts/consents to participate in the study if approved by PI.
2. Continues to be medically healthy and with clinically normal laboratory profiles, vital signs, and electrocardiograms (ECGs), in the opinion of the Investigator, assessed at Visit 1.
3. Is able to read and understand the Informed Consent Form (ICF).
4. Has signed the ICF.
5. Is willing and able to attend study appointments within specified time windows.
6. Is a female of childbearing potential (FOCP) who is either sexually inactive (abstinent) or, if sexually active, agrees to use one of the following acceptable birth control methods beginning at least 30 days prior to the first dose of SM and throughout the study:

   1. Simultaneous use of male condom and intra-uterine contraceptive device placed at least 4 weeks prior to first SM administration
   2. Surgically sterile male partner
   3. Simultaneous use of male condom and diaphragm with spermicide
   4. Established hormonal contraceptive

   Females are considered not to be of childbearing potential if they are either post-menopausal (amenorrhea for at least 2 years and serum follicle stimulating hormone [FSH] level of >40 IU/L) or permanently sterilized (e.g., bilateral tubal ligation, hysterectomy, bilateral oophorectomy for 6 months minimum prior to their Visit 1).
7. Is a male who:

   1. Agrees to use 2 methods of contraception in combination if his female partner is of childbearing potential; this combination of contraceptive methods must be used from Visit 1 to ≥ 1 month after the last dose of SM, OR
   2. Has been surgically sterilized prior to Visit 1.

Exclusion Criteria "A"

1. Is currently participating in another clinical trial other than Study 812P306.
2. Has any current psychiatric disorder per Diagnostic and Statistical Manual of Mental Disorders - 5th Edition (DSM-5) criteria other than ADHD with the following exceptions: ADHD is primary diagnosis with comorbidity/secondary diagnoses of major depression disorder (MDD), nicotine dependence, social anxiety disorder, generalized anxiety disorder, or phobias.
3. Current diagnosis of significant systemic disease and/or of a major psychiatric or neurological disorder, including history or family history of seizures or seizure-like disorders.
4. Current evidence of suicidality (suicidal thoughts or behaviors).
5. Female subjects who are pregnant, lactating and/or sexually active and not agreeing to use one of the acceptable birth control methods throughout the study.
6. Has a positive result on urine drug screen at Visit 1.
7. Use of prohibited concomitant medications including known CYP1A2 substrates (e.g., theophylline, melatonin) at the Visit 1 for the duration of the study.
8. Has a clinical laboratory value, vital sign value or ECG result at Visit 1 that is considered to be clinically significant in the opinion of the Investigator.
9. Has one or more clinical laboratory test values outside the reference range at Visit 1 that, in the opinion of the Investigator, are clinically significant, or any of the following (see Note below):

   * Serum creatinine > 1.5 times the upper limit of normal (ULN);
   * Serum total bilirubin > 1.5 times ULN;
   * Serum alanine aminotransferase or aspartate aminotransferase > 2 times ULN.
10. Has any of the following cardiology findings at Visit 1 (see Note below):

    * Abnormal ECG that is, in the Investigator's opinion, clinically significant;
    * PR interval > 220 ms;
    * QRS interval > 130 ms;
    * QTcF interval > 450 ms (for men) or > 470 ms (for women) (QT corrected using Fridericia's method);
    * Second- or third-degree atrioventricular block;
    * Any rhythm, other than sinus rhythm, that is interpreted by the Investigator to be clinically significant.
11. Any reason that, in the opinion of the Investigator, would prevent the subject from participating in the study.

Inclusion Criteria "B"

1. Is male or female, aged 18 to ≤ 65 years at screening.
2. Is able to read and understand the Informed Consent Form (ICF).
3. Written informed consent obtained from the subject (a signed ICF).
4. Weight within the normal or overweight ranges according to accepted values of the Body Mass Index (BMI) Chart (18.0 to 35.0 kg/m2).
5. Is able to swallow capsules whole, without crushing, chewing or cutting.
6. Is willing and able to attend study appointments within the specified time windows.
7. Has a primary diagnosis of ADHD according to the DSM-5 classification, with diagnosis made at least 6 months prior to screening and confirmed with Structured Clinical Interview for DSM-5 Clinical Trials version (SCID-5-CT; de novo subjects).
8. Has an AISRS total score of ≥ 24 at the screening (Visit 'S').
9. Has a CGI-S score of ≥ 4 (mildly ill or worse) at the screening (Visit 'S').
10. Females of childbearing potential (FOCP) must be either sexually inactive (abstinent) or, if sexually active, must agree to use one of the following acceptable birth control methods beginning at least 28 days prior to the first dose of SM and throughout the study:

    1. Simultaneous use of male condom and intra-uterine contraceptive device placed at least 4 weeks prior to first SM administration
    2. Surgically sterile male partner
    3. Simultaneous use of male condom and diaphragm with spermicide
    4. Established hormonal contraceptive

    Females are considered not to be of childbearing potential if they are either postmenopausal (amenorrhea for at least 2 years and serum follicle stimulating hormone [FSH] level of >40 IU/L) or permanently sterilized (e.g., bilateral tubal ligation, hysterectomy, bilateral oophorectomy for 6 months minimum prior to screening).
11. Males must:

    1. Use 2 methods of contraception in combination if his female partner is of childbearing potential; this combination of contraceptive methods must be used from Visit 1 (baseline) to ≥ 1 month after the last dose of SM; or
    2. Have been surgically sterilized prior to the Screening Visit.

Exclusion Criteria "B"

1. Is currently participating in another clinical trial or has participated in a clinical trial within 60 days prior screening, with the exception of Study 812P306.
2. Is a member of the study personnel or of their immediate families, or is a subordinate (or immediate family member of a subordinate) to any of the study personnel.
3. Female subjects who are pregnant, lactating and/or sexually active and not agreeing to use one of the acceptable birth control methods throughout the study.
4. Has a history of severe drug allergy or hypersensitivity, or known hypersensitivity, to the study medication.
5. Has a history of moderate or severe head trauma or other neurological disorder or systemic medical disease that, in the Investigator's opinion, is likely to affect central nervous system functioning. This would include subjects with:

   1. A current diagnosis of a major neurological disorder; or
   2. Seizures, seizure disorder or seizure-like events; or a history of seizure disorder within the immediate family (siblings, parents); or Encephalopathy
6. Has any history of schizophrenia, schizoaffective disorder, bipolar disorder, borderline personality disorder, antisocial personality disorder, narcissistic personality disorder, autism, post-traumatic stress disorder or obsessive-compulsive disorder.
7. Has any current psychiatric disorder (per DSM-5 criteria) other than ADHD with the following exceptions: ADHD is primary diagnoses with comorbidity/secondary diagnoses of major depression disorder (MDD), nicotine dependence, social anxiety disorder, generalized anxiety disorder, or phobias, and subject is not receiving pharmacological treatment for the comorbidity/secondary diagnoses (e.g., antidepressant for MDD) at time of screening nor for the duration of study.
8. Has organic mental disorders, or mental disorders due to a general medical condition (per DSM-5 criteria).
9. Has a current diagnosis or history of substance use disorder including alcohol use disorder (excluding nicotine and caffeine) (per DSM-5 criteria) within the 12 months prior to screening; or is assessed by the Investigator as having regularly consumed alcohol exceeding 21 units for males and 14 units for females per week (1 unit equals 340 mL of beer, 115 mL of wine, or 43 mL of spirits) within the 12 months prior to screening.
10. Is currently using, or has a positive result on the drug screening at the Screening Visit for drugs of abuse (alcohol, opiates, methadone, cocaine, methamphetamine [including ecstasy], phencyclidine, propoxyphene, methylphenidate, barbiturates, and benzodiazepines). If subject's serum drug screen for ethanol is positive at screening (Visit 'S') and the investigator determines subject does not have alcohol use disorder, then the subject may have a repeat serum drug screen for ethanol performed before Visit 1 within the allotted screening period (results must be received prior to Visit 1). If second serum drug screen for ethanol is positive, subject is excluded from participating in the study, however, if second serum drug screen for ethanol is negative, subject may proceed to Visit 1.
11. Is a (known or self-identified) current habitual/chronic cannabis user (medicinal or recreational); or

    * Has a positive urine drug screen for cannabis at screening (Visit 'S') and is considered, per the Investigator's judgement, to be a habitual/chronic cannabis user; or
    * Has a positive urine drug screen for cannabis at both the screening (Visit 'S') and follow-up drug screen (Visit 1), even though the subject is not considered, per the Investigator's judgement, to be a habitual/chronic cannabis user.

    Note: Subjects who have a positive urine drug screen for cannabis at screening (Visit 'S') but who are not considered, per the Investigator's judgement, to be a habitual/chronic cannabis user may, with Sponsor approval, undergo an additional urine drug screen at least 4 weeks after the initial urine drug screen at Visit 1 prior to randomization. Subjects must agree to refrain from cannabis use throughout study.
12. Has treatment-resistant ADHD based on a history of receipt of >2 approved ADHD medications that failed to adequately improve the subject's symptoms, with the exception of subjects who completed Study 812P306. A subject who is naïve to ADHD treatment is not excluded from study participation.
13. Has any other disorder for which its treatment takes priority over treatment of ADHD or is likely to interfere with study treatment, impair treatment compliance, or interfere with interpretation of study results.
14. Has a history of cancer, other than basal cell or Stage 1 squamous cell carcinoma of the skin that has not been in remission for > 5 years prior to the first dose of SM.
15. Has or has had one or more of the following conditions considered clinically significant/relevant by the Investigator in the context of the study:

    * cardiovascular disease
    * congestive heart failure
    * cardiac hypertrophy
    * arrhythmia
    * bradycardia (pulse < 50 bpm)
    * tachycardia (pulse > 100 bpm)
    * respiratory disease
    * hepatic impairment or renal insufficiency
    * metabolic disorder
    * endocrine disorder
    * gastrointestinal disorder
    * hematological disorder
    * infectious disorder
    * any clinically significant immunological condition
    * dermatological disorder
16. Exhibits clinically significant abnormal vital signs at screening (see Note below).
17. Has one or more screening clinical laboratory test values outside the reference range that, in the opinion of the Investigator, are clinically significant, or any of the following (see Note below):

    * Serum creatinine > 1.5 × the upper limit of normal (ULN);
    * Serum total bilirubin > 1.5 × ULN;
    * Serum alanine aminotransferase or aspartate aminotransferase > 2 × ULN.
18. Has any of the following cardiology findings at screening (see Note below):

    * Abnormal ECG that is, in the Investigator's opinion, clinically significant;
    * PR interval > 220 ms;
    * QRS interval > 130 ms;
    * QTcF interval > 450 ms (for men) or > 470 ms (for women) (QT corrected using Fridericia's method);
    * Second- or third-degree atrioventricular block;
    * Any rhythm, other than sinus rhythm, that is interpreted by the Investigator to be clinically significant.
19. Has any disease or medication that could, in the Investigator's opinion, interfere with the assessments of safety, tolerability, or efficacy, or interfere with study conduct or interpretation of results.
20. Evidence of infection with hepatitis B or C, or human immunodeficiency virus (HIV)-1 or HIV-2, as determined by results of testing at screening.
21. Lost or donated more than 450 mL of blood during the 30 days prior to screening.
22. Use of any investigational drug or prohibited concomitant medications including known CYP1A2 substrates (e.g., theophylline, melatonin) within 30 days or 5 halflives prior to Visit 1 (baseline) (whichever is longer) during the screening period or anticipated for the duration of the study.
23. History of unexplained loss of consciousness, unexplained syncope, unexplained irregular heartbeats or palpitations or near drowning with hospital admission.
24. Has attempted suicide within the 6 months prior to screening, or is at significant risk of suicide, either in the opinion of the Investigator or defined as a "yes" to suicidal ideation questions 4 or 5 or answering "yes" to suicidal behavior on the Columbia- Suicide Severity Rating Scale (C-SSRS) within the 6 months prior to screening.
25. In the Investigator's opinion, is unlikely to comply with the protocol or is unsuitable for any other reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rubin, MD, Study Director — Chief Medical Officer
Locations (38):
- United States (38):
  - South California Research LLC, Beverly Hills, California
  - Collaborative Neuroscience Network, Garden Grove, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California
  - Artemis Research Institue for Clinical Research, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Artemis Institute for Clinical Rearch, San Marcos, California
  - Collaborative Neuroscience Network LLC, Torrance, California
  - Gulfcoast Research Center, Fort Myers, Florida
  - Research Centers of America, Hollywood, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Meridien Research, Lakeland, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Clinical Neuroscience Solutions Inc., Orlando, Florida
  - CNS Healthcare, Orlando, Florida
  - Meridien Research, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - Psych Atlanta, Marietta, Georgia
  - Psychiatric Associates, Overland Park, Kansas
  - St. Charles Psychiatric Associates Midwest Research Center, Saint Charles, Missouri
  - Alivation Research, LLC, Lincoln, Nebraska
  - Altea Research Institute, Las Vegas, Nevada
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Hassmann Research Institute, Marlton, New Jersey
  - Princeton Medical Institute, Princeton, New Jersey
  - Bioscience Research, Mount Kisco, New York
  - The Medical Research Network LLC, New York, New York
  - Paradigm Research Professionals, Oklahoma City, Oklahoma
  - Clinical Neuroscience Solutions, Memphis, Tennessee
  - BioBehavioral Research of Austin P.C., Austin, Texas
  - FutureSearch Trials of Dallas, LLP, Dallas, Texas
  - Houston Clinical Trials, Houston, Texas
  - Family Psychiatry of the Woodlands, The Woodlands, Texas
  - Northwest Clinical Trials, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Childress A, Cutler AJ, Adler LA, Fry N, Asubonteng K, Maldonado-Cruz Z, Formella A, Rubin J. An Open-Label Extension Study Assessing the Long-Term Safety and Efficacy of Viloxazine Extended-Release Capsules in Adults with Attention-Deficit/Hyperactivity Disorder. CNS Drugs. 2024 Nov;38(11):891-907. doi: 10.1007/s40263-024-01120-0. Epub 2024 Oct 7. PMID 39373844

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open-Label Treatment
Started (Number of subjects "Started" is based on the Safety Population (defined as subjects who signed an Informed Consent and took at least one dose of SPN-812)) | 159
Not Treated (One subject signed Informed Consent and met eligibility criteria but did not dose, and four subjects signed Informed Consent but did not meet eligibility criteria.) | 5
Completed (Per protocol, a subject was considered as "Completed" if they either received 156 weeks of SPN-812 treatment or were discontinued prior to Week 156 due to SPN-812 being commercially available. All subjects considered "Completed" (n=26) were discontinued due to SPN-812 being commercially available prior to Week 156 (maximum SPN-812 exposure was 124 weeks).) | 26
Not Completed | 133
Not completed — Withdrawal by Subject | 42
Not completed — Adverse Event | 29
Not completed — Lost to Follow-up | 29
Not completed — Lack of Efficacy | 15
Not completed — Physician Decision | 1
Not completed — Non-Compliance With Study Drug | 6
Not completed — Other, Multiple Categories | 11

BASELINE CHARACTERISTICS:
Population: Baseline Participants is based on the Safety Population (defined as subjects who took at least one dose of SPN-812)
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (10.25)
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years of age | 119
  45 to 65 years of age | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31
  Not Hispanic or Latino | 128
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 133
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 159
Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The Adult ADHD Investigator Symptom Rating Scale (AISRS) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. It consists of 18 items that correspond to the 18 ADHD symptoms per the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). Each item is rated on a 4-point Likert-type scale from 0 (none) to 3 (severe). Total score = sum of 18 items (range: 0 to 54). The higher the score, the more severe the ADHD symptoms. Subjects who completed Study 812P306 (NCT04016779) were eligible to enroll in Study 812P311.
  units on a scale | 37.9 (6.34)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: The percent of subjects who took at least one dose of SPN-812 (Safety Population; N) and who reported at least one Adverse Event (n). The percent is calculated by dividing "the number of subjects who reported at least one Adverse Event (n)" by "the number of subjects in the Safety Population (N)" and multiplying the product by 100. The higher the percentage, the higher the incidence in the Safety Population
Time Frame: Up to 156 weeks
Population: Safety Population, defined as subjects who signed Informed Consent and took at least one dose of SPN-812.
Measure: Number; unit: percentage of subjects
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
percentage of subjects | 72.3

2. Secondary Outcome: The Effect of SPN-812 on Overall ADHD Symptoms as Measured by the Adult ADHD Investigator Symptom Rating Scale (AISRS)
Description: A secondary endpoint was the change from baseline in the Adult ADHD Investigator Symptom Rating Scale (AISRS) Total score by visit. The AISRS is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology in adults. The AISRS consists of 18 items that directly correspond to the 18 symptoms of ADHD per the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). The scale is subdivided into two subscales: Inattention (9 items) and Hyperactivity/Impulsivity (9 items). The clinician/investigator rates the subject on each item using a 4-point scale, where 0=none, 1=mild, 2=moderate, and 3=severe. The sum of the ratings of all 18 items yields the raw Total score (range: 0-54; the higher the Total score, the more severe the ADHD symptoms). Post-baseline raw Total scores are converted to a change from baseline Total score. A lower change from baseline AISRS Total Score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: Safety Population (N), defined as subjects who signed Informed Consent and took at least 1 dose of SPN-812. At each Visit/Week, data is summarized with descriptive statistics for the number of subjects analyzed (n; subjects with a valid AISRS assessment at baseline [pre-dosing] and at the respective post-baseline [after first dose] Visit/Week). Due to attrition and/or missing data, the number of subjects analyzed at each Visit/Week may be less than and unequal to Safety Population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
units on a scale
  Raw score; Baseline | 37.9 (6.34)
  Change from baseline score; Week 2: number analyzed (Participants) | 146
  Change from baseline score; Week 2 | -11.4 (9.50)
  Change from baseline score; Week 4: number analyzed (Participants) | 132
  Change from baseline score; Week 4 | -15.0 (10.13)
  Change from baseline score; Week 12: number analyzed (Participants) | 112
  Change from baseline score; Week 12 | -17.6 (10.69)
  Change from baseline score; Week 20: number analyzed (Participants) | 95
  Change from baseline score; Week 20 | -18.7 (11.46)
  Change from baseline score; Week 28: number analyzed (Participants) | 81
  Change from baseline score; Week 28 | -19.9 (9.88)
  Change from baseline score; Week 36: number analyzed (Participants) | 67
  Change from baseline score; Week 36 | -20.9 (10.39)
  Change from baseline score; Week 44: number analyzed (Participants) | 59
  Change from baseline score; Week 44 | -21.1 (10.27)
  Change from baseline score; Week 52: number analyzed (Participants) | 51
  Change from baseline score; Week 52 | -22.0 (10.40)
  Change from baseline score; Week 60: number analyzed (Participants) | 39
  Change from baseline score; Week 60 | -22.6 (11.34)
  Change from baseline score; Week 68: number analyzed (Participants) | 36
  Change from baseline score; Week 68 | -22.1 (11.32)
  Change from baseline score; Week 76: number analyzed (Participants) | 33
  Change from baseline score; Week 76 | -24.3 (10.64)
  Change from baseline score; Week 84: number analyzed (Participants) | 29
  Change from baseline score; Week 84 | -22.8 (10.86)
  Change from baseline score; Week 92: number analyzed (Participants) | 25
  Change from baseline score; Week 92 | -24.2 (11.94)
  Change from baseline score; Week 100: number analyzed (Participants) | 13
  Change from baseline score; Week 100 | -23.7 (11.72)
  Change from baseline score; Week 108: number analyzed (Participants) | 9
  Change from baseline score; Week 108 | -26.3 (11.29)
  Change from baseline score; Week 116: number analyzed (Participants) | 8
  Change from baseline score; Week 116 | -25.9 (12.41)
  Change from baseline score; Week 124: number analyzed (Participants) | 4
  Change from baseline score; Week 124 | -21.5 (16.26)

3. Secondary Outcome: The Effect of SPN-812 on Global Assessment of ADHD Symptom Severity as Measured by the Clinical Global Impression - Severity of Illness (CGI-S)
Description: An additional secondary endpoint was the change from baseline in the Clinical Global Impression - Severity of Illness (CGI-S) score at Week 6. The CGI-S is a single item clinician-rated assessment of the severity of subject's condition (ADHD symptoms) in relation to the clinician's total experience with patients with ADHD. The CGI-S is evaluated on a 7-point scale with 1 = Normal, not at all ill, asymptomatic, 2 = Borderline Ill, 3 = Mildly Ill, 4 = Moderately Ill, 5 = Markedly Ill, 6 = Severely Ill, and 7 = Among the most extremely ill patients (the higher the score, the more severe the overall ADHD symptoms). Post-baseline (raw) CGI-S scores are converted to a change from baseline score. A lower change from baseline CGI-S score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: Safety Population (N), defined as subjects who signed Informed Consent and took at least 1 dose of SPN-812. At each Visit/Week, data is summarized with descriptive statistics for the number of subjects analyzed (n; subjects with a valid CGI-S assessment at baseline [pre-dosing] and at the respective post-baseline [after first dose] Visit/Week). Due to attrition and/or missing data, the number of subjects analyzed at each Visit/Week may be less than and unequal to Safety Population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
units on a scale
  Raw score; Baseline | 4.6 (0.60)
  Change from baseline score; Week 2: number analyzed (Participants) | 146
  Change from baseline score; Week 2 | -1.0 (0.99)
  Change from baseline score; Week 4: number analyzed (Participants) | 132
  Change from baseline score; Week 4 | -1.3 (1.08)
  Change from baseline score; Week 12: number analyzed (Participants) | 112
  Change from baseline score; Week 12 | -1.6 (1.11)
  Change from baseline score; Week 20: number analyzed (Participants) | 95
  Change from baseline score; Week 20 | -1.8 (1.21)
  Change from baseline score; Week 28: number analyzed (Participants) | 81
  Change from baseline score; Week 28 | -1.8 (1.15)
  Change from baseline score; Week 36: number analyzed (Participants) | 67
  Change from baseline score; Week 36 | -2.0 (1.21)
  Change from baseline score; Week 44: number analyzed (Participants) | 59
  Change from baseline score; Week 44 | -2.0 (1.17)
  Change from baseline score; Week 52: number analyzed (Participants) | 51
  Change from baseline score; Week 52 | -2.1 (1.25)
  Change from baseline score; Week 60: number analyzed (Participants) | 39
  Change from baseline score; Week 60 | -2.2 (1.25)
  Change from baseline score; Week 68: number analyzed (Participants) | 36
  Change from baseline score; Week 68 | -2.1 (1.31)
  Change from baseline score; Week 76: number analyzed (Participants) | 33
  Change from baseline score; Week 76 | -2.4 (1.17)
  Change from baseline score; Week 84: number analyzed (Participants) | 29
  Change from baseline score; Week 84 | -2.3 (1.17)
  Change from baseline score; Week 92: number analyzed (Participants) | 25
  Change from baseline score; Week 92 | -2.5 (1.36)
  Change from baseline score; Week 100: number analyzed (Participants) | 13
  Change from baseline score; Week 100 | -2.3 (1.11)
  Change from baseline score; Week 108: number analyzed (Participants) | 9
  Change from baseline score; Week 108 | -2.7 (1.12)
  Change from baseline score; Week 116: number analyzed (Participants) | 8
  Change from baseline score; Week 116 | -2.4 (1.30)
  Change from baseline score; Week 124: number analyzed (Participants) | 4
  Change from baseline score; Week 124 | -1.5 (1.91)

4. Secondary Outcome: The Effect of SPN-812 on Clinical Global Impression - Severity of Illness (CGI-S) Responder Rate
Description: An additional secondary endpoint was the Clinical Global Impression - Severity of Illness (CGI-S) Responder Rate by visit. The CGI-S Responder Rate was defined as the percent of subjects with a CGI-S score of 1 or 2 ("responders"). The CGI-S is a single item clinician-rated assessment of the severity of subject's condition (ADHD symptoms) in relation to the clinician's total experience with patients with ADHD. The CGI-S is evaluated on a 7-point scale with 1 = Normal, not at all ill, asymptomatic, 2 = Borderline Ill, 3 = Mildly Ill, 4 = Moderately Ill, 5 = Markedly Ill, 6 = Severely Ill, and 7 = Among the most extremely ill patients. The responder rate (percent) is calculated by dividing "the number of 'responders' (m)" by "the number of subjects analyzed at the respective Visit/Week (n)" and multiplying the product by 100. Responder Rate values range from 0 to 100%. A percent >50% represents a greater number of "responders" versus "non-responders".
Time Frame: Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: Safety Population (N), defined as subjects who signed Informed Consent and took at least 1 dose of SPN-812. At each Visit/Week, percent is based on number of "responders" (m; CGI-S score of 1 or 2) and number of subjects analyzed (n; subjects with valid CGI-S assessment at baseline [pre-dosing] and at respective post-baseline [after first dose] Visit/Week). Due to attrition and/or missing data, the number of subjects analyzed at each Visit/Week may be less than and unequal to Safety Population.
Measure: Number; unit: percentage of subjects
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
percentage of subjects
  Percent of subjects; Week 2: number analyzed (Participants) | 146
  Percent of subjects; Week 2 | 16.4
  Percent of subjects; Week 4: number analyzed (Participants) | 132
  Percent of subjects; Week 4 | 23.5
  Percent of subjects; Week 12: number analyzed (Participants) | 112
  Percent of subjects; Week 12 | 29.5
  Percent of subjects; Week 20: number analyzed (Participants) | 95
  Percent of subjects; Week 20 | 36.8
  Percent of subjects; Week 28: number analyzed (Participants) | 81
  Percent of subjects; Week 28 | 42.0
  Percent of subjects; Week 36: number analyzed (Participants) | 67
  Percent of subjects; Week 36 | 47.8
  Percent of subjects; Week 44: number analyzed (Participants) | 59
  Percent of subjects; Week 44 | 42.4
  Percent of subjects; Week 52: number analyzed (Participants) | 51
  Percent of subjects; Week 52 | 56.9
  Percent of subjects; Week 60: number analyzed (Participants) | 39
  Percent of subjects; Week 60 | 53.8
  Percent of subjects; Week 68: number analyzed (Participants) | 36
  Percent of subjects; Week 68 | 52.8
  Percent of subjects; Week 76: number analyzed (Participants) | 33
  Percent of subjects; Week 76 | 60.6
  Percent of subjects; Week 84: number analyzed (Participants) | 29
  Percent of subjects; Week 84 | 55.2
  Percent of subjects; Week 92: number analyzed (Participants) | 25
  Percent of subjects; Week 92 | 68.0
  Percent of subjects; Week 100: number analyzed (Participants) | 13
  Percent of subjects; Week 100 | 61.5
  Percent of subjects; Week 108: number analyzed (Participants) | 9
  Percent of subjects; Week 108 | 66.7
  Percent of subjects; Week 116: number analyzed (Participants) | 8
  Percent of subjects; Week 116 | 62.5
  Percent of subjects; Week 124: number analyzed (Participants) | 4
  Percent of subjects; Week 124 | 25.0

5. Secondary Outcome: The Effect of SPN-812 on Global Assessment of Improvement of ADHD Symptoms as Measured by the Clinical Global Impression - Improvement Scale (CGI-I) Scale
Description: An additional secondary endpoint was the Clinical Global Impression - Improvement (CGI-I) score by visit. The CGI-I scale is a single item clinician-rated assessment of how much the subject's condition (ADHD) has improved, worsened or has not changed relative to his/her baseline state prior to the beginning of treatment. The CGI-I is rated on a 7-point scale from 1 to 7, where 1 = "very much improved", 2 = "much improved", 3 = "minimally improved", 4 = "no change", 5 = "minimally worse", 6 = "much worse", and 7 = "very much worse". A CGI-I score <4 represents a better outcome.
Time Frame: Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: Safety Population (N), defined as subjects who signed Informed Consent and took at least 1 dose of SPN-812. At each Visit/Week, data is summarized with descriptive statistics for the total number of subjects analyzed (n; subjects with a valid CGI-I assessment at the respective post-baseline [after first dose] Visit/Week). Due to attrition and/or missing data, the number of subjects analyzed at each Visit/Week may be less than and unequal to Safety Population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
units on a scale
  Score; Week 2: number analyzed (Participants) | 146
  Score; Week 2 | 2.9 (0.96)
  Score; Week 4: number analyzed (Participants) | 132
  Score; Week 4 | 2.6 (0.97)
  Score; Week 12: number analyzed (Participants) | 112
  Score; Week 12 | 2.4 (1.02)
  Score; Week 20: number analyzed (Participants) | 95
  Score; Week 20 | 2.2 (1.00)
  Score; Week 28: number analyzed (Participants) | 81
  Score; Week 28 | 2.2 (0.93)
  Score; Week 36: number analyzed (Participants) | 67
  Score; Week 36 | 1.9 (0.93)
  Score; Week 44: number analyzed (Participants) | 59
  Score; Week 44 | 1.9 (0.88)
  Score; Week 52: number analyzed (Participants) | 51
  Score; Week 52 | 1.9 (1.12)
  Score; Week 60: number analyzed (Participants) | 39
  Score; Week 60 | 1.8 (0.87)
  Score; Week 68: number analyzed (Participants) | 36
  Score; Week 68 | 1.8 (0.97)
  Score; Week 76: number analyzed (Participants) | 33
  Score; Week 76 | 1.8 (0.85)
  Score; Week 84: number analyzed (Participants) | 29
  Score; Week 84 | 1.9 (0.88)
  Score; Week 92: number analyzed (Participants) | 25
  Score; Week 92 | 1.8 (1.03)
  Score; Week 100: number analyzed (Participants) | 13
  Score; Week 100 | 1.8 (0.90)
  Score; Week 108: number analyzed (Participants) | 9
  Score; Week 108 | 1.7 (0.71)
  Score; Week 116: number analyzed (Participants) | 8
  Score; Week 116 | 1.8 (0.71)
  Score; Week 124: number analyzed (Participants) | 4
  Score; Week 124 | 2.5 (1.29)

6. Secondary Outcome: The Effect of SPN-812 on Clinical Global Impression - Improvement (CGI-I) Responder Rate
Description: An additional endpoint was Clinical Global Impression - Improvement (CGI-I) Responder Rate by visit. The CGI-I Responder Rate was defined as the percent of subjects with a CGI-I score of 1 or 2 ("responders"). The CGI-I scale is a single item clinician-rated assessment of how much the subject's condition (ADHD) has improved, worsened or has not changed relative to his/her baseline state prior to the beginning of treatment. The CGI-I is rated on a 7-point scale from 1 to 7, where 1 = "very much improved", 2 = "much improved", 3 = "minimally improved", 4 = "no change", 5 = "minimally worse", 6 = "much worse", and 7 = "very much worse". The responder rate (percent) is calculated by dividing "the number of 'responders' (m)" by "the number of subjects analyzed at the respective Visit/Week (n)" and multiplying the product by 100. Responder Rate values range from 0 to 100%. A percent >50% represents a greater number of "responders" versus "non-responders".
Time Frame: Weeks 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: Safety Population (N), defined as subjects who signed Informed Consent and took at least 1 dose of SPN-812. At each Visit/Week, the percent is based on number of "responders" (m; CGI-I score of 1 or 2) and number of subjects analyzed (n; subjects with a valid CGI-I assessment at respective post-baseline [after first dose] Visit/Week). Due to attrition and/or missing data, the number of subjects analyzed at each Visit/Week may be less than and unequal to Safety Population.
Measure: Number; unit: percentage of subjects
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
percentage of subjects
  Percent of subjects; Week 2: number analyzed (Participants) | 146
  Percent of subjects; Week 2 | 32.9
  Percent of subjects; Week 4: number analyzed (Participants) | 132
  Percent of subjects; Week 4 | 47.7
  Percent of subjects; Week 12: number analyzed (Participants) | 112
  Percent of subjects; Week 12 | 61.6
  Percent of subjects; Week 20: number analyzed (Participants) | 95
  Percent of subjects; Week 20 | 68.4
  Percent of subjects; Week 28: number analyzed (Participants) | 81
  Percent of subjects; Week 28 | 70.4
  Percent of subjects; Week 36: number analyzed (Participants) | 67
  Percent of subjects; Week 36 | 76.1
  Percent of subjects; Week 44: number analyzed (Participants) | 59
  Percent of subjects; Week 44 | 79.7
  Percent of subjects; Week 52: number analyzed (Participants) | 51
  Percent of subjects; Week 52 | 80.4
  Percent of subjects; Week 60: number analyzed (Participants) | 39
  Percent of subjects; Week 60 | 84.6
  Percent of subjects; Week 68: number analyzed (Participants) | 36
  Percent of subjects; Week 68 | 77.8
  Percent of subjects; Week 76: number analyzed (Participants) | 33
  Percent of subjects; Week 76 | 84.8
  Percent of subjects; Week 84: number analyzed (Participants) | 29
  Percent of subjects; Week 84 | 82.8
  Percent of subjects; Week 92: number analyzed (Participants) | 25
  Percent of subjects; Week 92 | 80.0
  Percent of subjects; Week 100: number analyzed (Participants) | 13
  Percent of subjects; Week 100 | 84.6
  Percent of subjects; Week 108: number analyzed (Participants) | 9
  Percent of subjects; Week 108 | 88.9
  Percent of subjects; Week 116: number analyzed (Participants) | 8
  Percent of subjects; Week 116 | 87.5
  Percent of subjects; Week 124: number analyzed (Participants) | 4
  Percent of subjects; Week 124 | 50.0

7. Secondary Outcome: Effect of SPN-812 on Symptoms of Anxiety as Measured by the Generalized Anxiety Disorder 7-Item (GAD-7) Scale
Description: An additional secondary endpoint was the change from baseline in the Generalized Anxiety Disorder 7-Item (GAD-7) Total Score by visit. The GAD-7 is a self-reported 7-item questionnaire for screening and measuring the severity of generalized anxiety disorder. The subject rates each item on 4-point scale (0-3), where 0 = "Not at all", 1 = "Several days", 2 = "Over half the days", and 3 = "Nearly every day". The sum of the 7 items yields a raw GAD-7 Total score (range between 0 to 21); the higher the GAD-7 Total score, the more severe the symptoms of anxiety. Post-baseline raw GAD-7 Total scores are converted to a change from baseline score. A lower change from baseline GAD-7 Total score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: Safety Population (N), defined as subjects who signed Informed Consent and took at least 1 dose of SPN-812. At each Visit/Week, data is summarized with descriptive statistics for the number of subjects analyzed (n; subjects with a valid GAD-7 assessment at baseline [pre-dosing] and at the respective post-baseline [after first dose] Visit/Week). Due to attrition and/or missing data, the number of subjects analyzed at each Visit/Week may be less than and unequal to Safety Population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
units on a scale
  Raw score; Baseline: number analyzed (Participants) | 158
  Raw score; Baseline | 5.9 (4.47)
  Change from baseline score; Week 2: number analyzed (Participants) | 142
  Change from baseline score; Week 2 | -1.2 (3.93)
  Change from baseline score; Week 4: number analyzed (Participants) | 131
  Change from baseline score; Week 4 | -1.6 (4.40)
  Change from baseline score; Week 12: number analyzed (Participants) | 110
  Change from baseline score; Week 12 | -1.7 (4.63)
  Change from baseline score; Week 20: number analyzed (Participants) | 94
  Change from baseline score; Week 20 | -2.0 (3.99)
  Change from baseline score; Week 28: number analyzed (Participants) | 80
  Change from baseline score; Week 28 | -2.0 (3.90)
  Change from baseline score; Week 36: number analyzed (Participants) | 67
  Change from baseline score; Week 36 | -1.3 (4.43)
  Change from baseline score; Week 44: number analyzed (Participants) | 59
  Change from baseline score; Week 44 | -2.1 (3.50)
  Change from baseline score; Week 52: number analyzed (Participants) | 51
  Change from baseline score; Week 52 | -2.0 (4.25)
  Change from baseline score; Week 60: number analyzed (Participants) | 38
  Change from baseline score; Week 60 | -1.7 (3.87)
  Change from baseline score; Week 68: number analyzed (Participants) | 36
  Change from baseline score; Week 68 | -2.4 (3.87)
  Change from baseline score; Week 76: number analyzed (Participants) | 33
  Change from baseline score; Week 76 | -2.6 (3.41)
  Change from baseline score; Week 84: number analyzed (Participants) | 28
  Change from baseline score; Week 84 | -2.4 (4.04)
  Change from baseline score; Week 92: number analyzed (Participants) | 25
  Change from baseline score; Week 92 | -3.2 (3.40)
  Change from baseline score; Week 100: number analyzed (Participants) | 13
  Change from baseline score; Week 100 | -3.2 (3.74)
  Change from baseline score; Week 108: number analyzed (Participants) | 9
  Change from baseline score; Week 108 | -3.1 (4.14)
  Change from baseline score; Week 116: number analyzed (Participants) | 8
  Change from baseline score; Week 116 | -3.5 (4.00)
  Change from baseline score; Week 124: number analyzed (Participants) | 4
  Change from baseline score; Week 124 | -3.8 (5.56)

8. Secondary Outcome: Effect of SPN-812 on Hyperactivity/Impulsivity (H/I) Symptoms as Measured by the Adult ADHD Investigator Symptom Rating H/I Subscale
Description: An additional secondary endpoint was the change from baseline in the Adult ADHD Investigator Symptom Rating Scale (AISRS) "Hyperactivity/Impulsivity" (H/I) subscale score. The AISRS is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology in adults. The AISRS consists of 18 items that directly correspond to the 18 symptoms of ADHD per the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). The scale is subdivided into two subscales: Inattention (9 items) and H/I (9 items). The clinician/investigator rates the subject on each item using a 4-point scale, where 0=none, 1=mild, 2=moderate, and 3=severe. The sum of the nine H/I items yields the raw H/I subscale score (range: 0-27; the higher the H/I subscale score, the more severe the H/I symptoms). Post-baseline raw H/I subscale scores are converted to a change from baseline score. A lower change from baseline H/I subscale score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: Safety Population (N), defined as subjects who signed Informed Consent and took at least 1 dose of SPN-812. At each Visit/Week, data is summarized with descriptive statistics for the number of subjects analyzed (n; subjects with a valid AISRS assessment at baseline [pre-dosing] and at the respective post-baseline [after first dose] Visit/Week). Due to attrition and/or missing data, the number of subjects analyzed at each Visit/Week may be less than and unequal to the Safety Population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
units on a scale
  Raw score; Baseline | 16.2 (4.92)
  Change from baseline score; Week 2: number analyzed (Participants) | 146
  Change from baseline score; Week 2 | -5.3 (5.35)
  Change from baseline score; Week 4: number analyzed (Participants) | 132
  Change from baseline score; Week 4 | -7.1 (5.27)
  Change from baseline score; Week 12: number analyzed (Participants) | 112
  Change from baseline score; Week 12 | -8.1 (5.67)
  Change from baseline score; Week 20: number analyzed (Participants) | 95
  Change from baseline score; Week 20 | -8.4 (5.83)
  Change from baseline score; Week 28: number analyzed (Participants) | 81
  Change from baseline score; Week 28 | -8.7 (5.30)
  Change from baseline score; Week 36: number analyzed (Participants) | 67
  Change from baseline score; Week 36 | -9.7 (5.80)
  Change from baseline score; Week 44: number analyzed (Participants) | 59
  Change from baseline score; Week 44 | -10.1 (5.28)
  Change from baseline score; Week 52: number analyzed (Participants) | 51
  Change from baseline score; Week 52 | -10.2 (5.84)
  Change from baseline score; Week 60: number analyzed (Participants) | 39
  Change from baseline score; Week 60 | -10.1 (5.96)
  Change from baseline score; Week 68: number analyzed (Participants) | 36
  Change from baseline score; Week 68 | -10.4 (5.52)
  Change from baseline score; Week 76: number analyzed (Participants) | 33
  Change from baseline score; Week 76 | -11.1 (5.31)
  Change from baseline score; Week 84: number analyzed (Participants) | 29
  Change from baseline score; Week 84 | -10.5 (5.42)
  Change from baseline score; Week 92: number analyzed (Participants) | 25
  Change from baseline score; Week 92 | -11.1 (5.34)
  Change from baseline score; Week 100: number analyzed (Participants) | 13
  Change from baseline score; Week 100 | -11.1 (5.25)
  Change from baseline score; Week 108: number analyzed (Participants) | 9
  Change from baseline score; Week 108 | -12.2 (4.94)
  Change from baseline score; Week 116: number analyzed (Participants) | 8
  Change from baseline score; Week 116 | -11.9 (4.97)
  Change from baseline score; Week 124: number analyzed (Participants) | 4
  Change from baseline score; Week 124 | -10.3 (7.93)

9. Secondary Outcome: Effect of SPN-812 on Inattention (IA) Symptoms as Measured by the Adult ADHD Investigator Symptom Rating IA Subscale
Description: An additional secondary endpoint was the change from baseline in the Adult ADHD Investigator Symptom Rating Scale (AISRS) "Inattention" (IA) subscale score. The AISRS is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology in adults. The AISRS consists of 18 items that directly correspond to the 18 symptoms of ADHD per the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). The scale is subdivided into two subscales: Inattention (9 items) and Hyperactivity/Impulsivity (9 items). The clinician/investigator rates the subject on each item using a 4-point scale, where 0=none, 1=mild, 2=moderate, and 3=severe. The sum of the nine IA items yields the raw IA subscale score (range: 0-27; the higher the IA subscale score, the more severe the IA symptoms). Post-baseline raw IA subscale scores are converted to a change from baseline score. A lower change from baseline IA subscale score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
units on a scale
  Raw score; Baseline | 21.6 (3.39)
  Change from baseline score; Week 2: number analyzed (Participants) | 146
  Change from baseline score; Week 2 | -6.1 (5.58)
  Change from baseline score; Week 4: number analyzed (Participants) | 132
  Change from baseline score; Week 4 | -7.9 (6.11)
  Change from baseline score; Week 12: number analyzed (Participants) | 112
  Change from baseline score; Week 12 | -9.5 (6.26)
  Change from baseline score; Week 20: number analyzed (Participants) | 95
  Change from baseline score; Week 20 | -10.2 (6.99)
  Change from baseline score; Week 28: number analyzed (Participants) | 81
  Change from baseline score; Week 28 | -11.2 (5.91)
  Change from baseline score; Week 36: number analyzed (Participants) | 67
  Change from baseline score; Week 36 | -11.3 (5.94)
  Change from baseline score; Week 44: number analyzed (Participants) | 59
  Change from baseline score; Week 44 | -10.9 (6.56)
  Change from baseline score; Week 52: number analyzed (Participants) | 51
  Change from baseline score; Week 52 | -11.8 (6.00)
  Change from baseline score; Week 60: number analyzed (Participants) | 39
  Change from baseline score; Week 60 | -12.5 (6.63)
  Change from baseline score; Week 68: number analyzed (Participants) | 36
  Change from baseline score; Week 68 | -11.6 (7.06)
  Change from baseline score; Week 76: number analyzed (Participants) | 33
  Change from baseline score; Week 76 | -13.2 (6.31)
  Change from baseline score; Week 84: number analyzed (Participants) | 29
  Change from baseline score; Week 84 | -12.2 (6.94)
  Change from baseline score; Week 92: number analyzed (Participants) | 25
  Change from baseline score; Week 92 | -13.2 (7.36)
  Change from baseline score; Week 100: number analyzed (Participants) | 13
  Change from baseline score; Week 100 | -12.6 (6.89)
  Change from baseline score; Week 108: number analyzed (Participants) | 9
  Change from baseline score; Week 108 | -14.1 (7.18)
  Change from baseline score; Week 116: number analyzed (Participants) | 8
  Change from baseline score; Week 116 | -14.0 (8.14)
  Change from baseline score; Week 124: number analyzed (Participants) | 4
  Change from baseline score; Week 124 | -11.3 (8.54)

10. Secondary Outcome: Effect of SPN-812 on the 50% Adult ADHD Investigator Symptom Rating Scale (AISRS) Responder Rate
Description: An additional secondary endpoint was the 50% Adult ADHD Investigator Symptom Rating Scale (AISRS) Responder Rate by visit. The AISRS is an ADHD-specific rating scale designed/validated to assess the 18 symptoms (items) of ADHD per the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). Each item is rated on a 4-point scale (0=none, 1=mild, 2=moderate, 3=severe). The sum of the 18 ratings yields the Total score (range: 0-54; higher score represents severer symptoms). Percent reduction is calculated for each post-baseline AISRS score: [("Post-baseline" - "Baseline")/"Baseline"] x 100; range: 0 to 100%; a "responder" is a subject with a 50% or greater reduction in change from baseline Total score. Responder rate (percent of responders) is calculated: ["number of 'responders' (m)" / "number of subjects analyzed" (n)] X 100; range: 0 to 100%. A Responder Rate greater than 50%, represents more "responders" versus "nonresponders".
Time Frame: Weeks 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: Safety Population (N), defined as subjects who signed Informed Consent and took at least 1 dose of SPN-812. At each Visit/Week, the percent is based on number of "responders" (m) and number of subjects analyzed (n; subjects with a valid AISRS assessment at baseline [pre-dosing] and at respective post-baseline [after first dose] Visit/Week). Due to attrition and/or missing data, the number of subjects analyzed at each Visit/Week may be less than and unequal to Safety Population.
Measure: Number; unit: percentage of subjects
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
percentage of subjects
  Percent of subjects; Week 2: number analyzed (Participants) | 146
  Percent of subjects; Week 2 | 22.6
  Percent of subjects; Week 4: number analyzed (Participants) | 132
  Percent of subjects; Week 4 | 38.6
  Percent of subjects; Week 12: number analyzed (Participants) | 112
  Percent of subjects; Week 12 | 58.0
  Percent of subjects; Week 20: number analyzed (Participants) | 95
  Percent of subjects; Week 20 | 55.8
  Percent of subjects; Week 28: number analyzed (Participants) | 81
  Percent of subjects; Week 28 | 61.7
  Percent of subjects; Week 36: number analyzed (Participants) | 67
  Percent of subjects; Week 36 | 64.2
  Percent of subjects; Week 44: number analyzed (Participants) | 59
  Percent of subjects; Week 44 | 64.4
  Percent of subjects; Week 52: number analyzed (Participants) | 51
  Percent of subjects; Week 52 | 66.7
  Percent of subjects; Week 60: number analyzed (Participants) | 39
  Percent of subjects; Week 60 | 71.8
  Percent of subjects; Week 68: number analyzed (Participants) | 36
  Percent of subjects; Week 68 | 63.9
  Percent of subjects; Week 76: number analyzed (Participants) | 33
  Percent of subjects; Week 76 | 78.8
  Percent of subjects; Week 84: number analyzed (Participants) | 29
  Percent of subjects; Week 84 | 72.4
  Percent of subjects; Week 92: number analyzed (Participants) | 25
  Percent of subjects; Week 92 | 80.0
  Percent of subjects; Week 100: number analyzed (Participants) | 13
  Percent of subjects; Week 100 | 69.2
  Percent of subjects; Week 108: number analyzed (Participants) | 9
  Percent of subjects; Week 108 | 77.8
  Percent of subjects; Week 116: number analyzed (Participants) | 8
  Percent of subjects; Week 116 | 75.0
  Percent of subjects; Week 124: number analyzed (Participants) | 4
  Percent of subjects; Week 124 | 50.0

11. Secondary Outcome: Effect of SPN-812 on the 30% Adult ADHD Investigator Symptom Rating Scale (AISRS) Responder Rate
Description: An additional secondary endpoint was the 30% Adult ADHD Investigator Symptom Rating Scale (AISRS) Responder Rate by visit. The AISRS is an ADHD-specific rating scale designed/validated to assess the 18 symptoms (items) of ADHD per the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). Each item is rated on a 4-point scale (0=none, 1=mild, 2=moderate, 3=severe). The sum of the 18 ratings yields the Total score (range: 0-54; higher score represents severer symptoms). Percent reduction is calculated for each post-baseline AISRS score: [("Post-baseline" - "Baseline")/"Baseline"] x 100; range: 0 to 100%; a "responder" is a subject with a 50% or greater reduction in change from baseline Total score. Responder rate (percent of responders) is calculated: ["number of 'responders' (m)" / "number of subjects analyzed" (n)] X 100; range: 0 to 100%. A Responder Rate greater than 30%, represents more "responders" versus "nonresponders".
Time Frame: Weeks 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 10
Measure: Number; unit: percentage of subjects
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
percentage of subjects
  Percent of subjects; Week 2: number analyzed (Participants) | 146
  Percent of subjects; Week 2 | 46.6
  Percent of subjects; Week 4: number analyzed (Participants) | 132
  Percent of subjects; Week 4 | 64.4
  Percent of subjects; Week 12: number analyzed (Participants) | 112
  Percent of subjects; Week 12 | 72.3
  Percent of subjects; Week 20: number analyzed (Participants) | 95
  Percent of subjects; Week 20 | 77.9
  Percent of subjects; Week 28: number analyzed (Participants) | 81
  Percent of subjects; Week 28 | 80.2
  Percent of subjects; Week 36: number analyzed (Participants) | 67
  Percent of subjects; Week 36 | 83.6
  Percent of subjects; Week 44: number analyzed (Participants) | 59
  Percent of subjects; Week 44 | 86.4
  Percent of subjects; Week 52: number analyzed (Participants) | 51
  Percent of subjects; Week 52 | 84.3
  Percent of subjects; Week 60: number analyzed (Participants) | 39
  Percent of subjects; Week 60 | 87.2
  Percent of subjects; Week 68: number analyzed (Participants) | 36
  Percent of subjects; Week 68 | 91.7
  Percent of subjects; Week 76: number analyzed (Participants) | 33
  Percent of subjects; Week 76 | 93.9
  Percent of subjects; Week 84: number analyzed (Participants) | 29
  Percent of subjects; Week 84 | 89.7
  Percent of subjects; Week 92: number analyzed (Participants) | 25
  Percent of subjects; Week 92 | 92.0
  Percent of subjects; Week 100: number analyzed (Participants) | 13
  Percent of subjects; Week 100 | 92.3
  Percent of subjects; Week 108: number analyzed (Participants) | 9
  Percent of subjects; Week 108 | 88.9
  Percent of subjects; Week 116: number analyzed (Participants) | 8
  Percent of subjects; Week 116 | 87.5
  Percent of subjects; Week 124: number analyzed (Participants) | 4
  Percent of subjects; Week 124 | 75.0

12. Secondary Outcome: Effect of SPN-812 on Overall Executive Function in Adults With ADHD as Measured by the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A; Self Report)
Description: An additional secondary endpoint was the change from baseline in the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) Global Executive Composite (GEC) T-score by visit. The BRIEF-A is a 75-item self-rating scale that assesses overall functioning (GEC) and 9 non-overlapping scales among 2 summary index scales (Metacognition Index [MI] and Behavioral Regulation Index [BRI]) that assess aspects of executive function and problems with self-regulation from the perspective of the individual. Subjects rate each item on a 3-point scale (1=Never, 2=Sometimes, or 3=Often) based on their experience in past month. The sum of 70 items yields the GEC raw score (range: 70-210), which is converted to a T-score (normative population mean=50 and standard deviation=10; T-score ≥ 65 is considered abnormally elevated). Post-baseline GEC T-scores are converted to a change from baseline T-score. A lower change from baseline GEC T-score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: Safety Population (N), defined as subjects who signed Informed Consent and took at least 1 dose of SPN-812. At each Visit/Week, data is summarized with descriptive statistics for the number of subjects analyzed (n; subjects with a valid BRIEF-A assessment at baseline [pre-dosing] and at the respective post-baseline [after first dose] Visit/Week). Due to attrition and/or missing data, the number of subjects analyzed at each Visit/Week may be less than and unequal to Safety Population.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
T-score
  T-score; Baseline: number analyzed (Participants) | 156
  T-score; Baseline | 70.4 (10.94)
  Change from baseline T-score; Week 2: number analyzed (Participants) | 14
  Change from baseline T-score; Week 2 | -1.9 (8.20)
  Change from baseline T-score; Week 4: number analyzed (Participants) | 117
  Change from baseline T-score; Week 4 | -9.3 (9.91)
  Change from baseline T-score; Week 12: number analyzed (Participants) | 104
  Change from baseline T-score; Week 12 | -10.0 (11.46)
  Change from baseline T-score; Week 20: number analyzed (Participants) | 91
  Change from baseline T-score; Week 20 | -13.0 (12.20)
  Change from baseline T-score; Week 28: number analyzed (Participants) | 78
  Change from baseline T-score; Week 28 | -14.2 (12.76)
  Change from baseline T-score; Week 36: number analyzed (Participants) | 65
  Change from baseline T-score; Week 36 | -14.6 (12.00)
  Change from baseline T-score; Week 44: number analyzed (Participants) | 57
  Change from baseline T-score; Week 44 | -14.2 (11.72)
  Change from baseline T-score; Week 52: number analyzed (Participants) | 50
  Change from baseline T-score; Week 52 | -15.1 (13.84)
  Change from baseline T-score; Week 60: number analyzed (Participants) | 38
  Change from baseline T-score; Week 60 | -15.4 (14.32)
  Change from baseline T-score; Week 68: number analyzed (Participants) | 36
  Change from baseline T-score; Week 68 | -16.3 (15.21)
  Change from baseline T-score; Week 76: number analyzed (Participants) | 33
  Change from baseline T-score; Week 76 | -16.7 (15.10)
  Change from baseline T-score; Week 84: number analyzed (Participants) | 28
  Change from baseline T-score; Week 84 | -15.9 (12.72)
  Change from baseline T-score; Week 92: number analyzed (Participants) | 25
  Change from baseline T-score; Week 92 | -14.8 (15.00)
  Change from baseline T-score; Week 100: number analyzed (Participants) | 13
  Change from baseline T-score; Week 100 | -16.1 (16.27)
  Change from baseline T-score; Week 108: number analyzed (Participants) | 9
  Change from baseline T-score; Week 108 | -17.8 (20.60)
  Change from baseline T-score; Week 116: number analyzed (Participants) | 7
  Change from baseline T-score; Week 116 | -12.9 (17.28)
  Change from baseline T-score; Week 124: number analyzed (Participants) | 3
  Change from baseline T-score; Week 124 | -13.7 (28.54)

13. Secondary Outcome: Effect of SPN-812 on Behavior Regulation in Adults With ADHD as Measured by the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A; Self Report)
Description: An additional secondary endpoint was the change from baseline in the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) Behavioral Regulation Index (BRI) T-score by visit. The BRIEF-A is a 75-item self-rating scale that assesses overall functioning and 9 non-overlapping scales among 2 summary index scales. The BRI captures the ability to maintain appropriate regulatory control of one's own behavior and emotional responses. Subjects rate each item on a 3-point scale (1=Never, 2=Sometimes, or 3=Often) based on their experience in past month. The sum of 30 items yields the BRI raw score (range: 30-90), which is converted to a T-score (normative population mean=50 and standard deviation=10; T-score ≥ 65 is considered abnormally elevated). Post-baseline BRI T-scores are converted to a change from baseline T-score. A lower change from baseline BRI T-score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
T-score
  T-score; Baseline: number analyzed (Participants) | 157
  T-score; Baseline | 63.0 (11.16)
  Change from baseline T-score; Week 2: number analyzed (Participants) | 14
  Change from baseline T-score; Week 2 | -0.5 (5.92)
  Change from baseline T-score; Week 4: number analyzed (Participants) | 119
  Change from baseline T-score; Week 4 | -8.4 (9.32)
  Change from baseline T-score; Week 12: number analyzed (Participants) | 106
  Change from baseline T-score; Week 12 | -8.7 (10.66)
  Change from baseline T-score; Week 20: number analyzed (Participants) | 94
  Change from baseline T-score; Week 20 | -10.6 (10.70)
  Change from baseline T-score; Week 28: number analyzed (Participants) | 79
  Change from baseline T-score; Week 28 | -10.7 (11.59)
  Change from baseline T-score; Week 36: number analyzed (Participants) | 66
  Change from baseline T-score; Week 36 | -11.7 (10.86)
  Change from baseline T-score; Week 44: number analyzed (Participants) | 58
  Change from baseline T-score; Week 44 | -11.0 (10.61)
  Change from baseline T-score; Week 52: number analyzed (Participants) | 51
  Change from baseline T-score; Week 52 | -12.3 (12.88)
  Change from baseline T-score; Week 60: number analyzed (Participants) | 38
  Change from baseline T-score; Week 60 | -11.6 (13.09)
  Change from baseline T-score; Week 68: number analyzed (Participants) | 36
  Change from baseline T-score; Week 68 | -12.8 (14.04)
  Change from baseline T-score; Week 76: number analyzed (Participants) | 33
  Change from baseline T-score; Week 76 | -13.1 (13.43)
  Change from baseline T-score; Week 84: number analyzed (Participants) | 28
  Change from baseline T-score; Week 84 | -13.1 (10.66)
  Change from baseline T-score; Week 92: number analyzed (Participants) | 25
  Change from baseline T-score; Week 92 | -12.0 (11.82)
  Change from baseline T-score; Week 100: number analyzed (Participants) | 13
  Change from baseline T-score; Week 100 | -12.8 (12.10)
  Change from baseline T-score; Week 108: number analyzed (Participants) | 9
  Change from baseline T-score; Week 108 | -14.8 (18.40)
  Change from baseline T-score; Week 116: number analyzed (Participants) | 7
  Change from baseline T-score; Week 116 | -12.9 (15.69)
  Change from baseline T-score; Week 124: number analyzed (Participants) | 3
  Change from baseline T-score; Week 124 | -10.0 (24.56)

14. Secondary Outcome: Effect of SPN-812 on Metacognition in Adults With ADHD as Measured by the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A; Self Report)
Description: An additional secondary endpoint was the change from baseline in the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) Metacognition Index (MI) T-score. The BRIEF-A is a 75-item self-rating scale that assesses overall functioning and 9 non-overlapping scales among 2 summary index scales. MI reflects individual's ability to problem solve (includes initiate activity, generate ideas, sustain working memory, plan/organize approaches, monitor success/failure, and organize materials/environment). Subjects rate each item on a 3-point scale (1=Never, 2=Sometimes, or 3=Often) based on their experience in past month. The sum of 40 items yields the MI raw score (range: 40-120), which is converted to a T-score (normative population mean=50 and standard deviation=10; T-score ≥ 65 is considered abnormally elevated). Post-baseline MI T-scores are converted to a change from baseline T-score. A lower change from baseline MI T-score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
T-score
  T-score; Baseline: number analyzed (Participants) | 156
  T-score; Baseline | 73.4 (11.56)
  Change from baseline T-score; Week 2: number analyzed (Participants) | 14
  Change from baseline T-score; Week 2 | -2.4 (9.36)
  Change from baseline T-score; Week 4: number analyzed (Participants) | 117
  Change from baseline T-score; Week 4 | -8.9 (10.45)
  Change from baseline T-score; Week 12: number analyzed (Participants) | 104
  Change from baseline T-score; Week 12 | -10.0 (11.80)
  Change from baseline T-score; Week 20: number analyzed (Participants) | 91
  Change from baseline T-score; Week 20 | -12.9 (13.00)
  Change from baseline T-score; Week 28: number analyzed (Participants) | 78
  Change from baseline T-score; Week 28 | -15.0 (13.04)
  Change from baseline T-score; Week 36: number analyzed (Participants) | 65
  Change from baseline T-score; Week 36 | -15.0 (12.46)
  Change from baseline T-score; Week 44: number analyzed (Participants) | 57
  Change from baseline T-score; Week 44 | -14.8 (12.02)
  Change from baseline T-score; Week 52: number analyzed (Participants) | 50
  Change from baseline T-score; Week 52 | -15.3 (13.58)
  Change from baseline T-score; Week 60: number analyzed (Participants) | 38
  Change from baseline T-score; Week 60 | -16.2 (14.24)
  Change from baseline T-score; Week 68: number analyzed (Participants) | 36
  Change from baseline T-score; Week 68 | -16.9 (15.32)
  Change from baseline T-score; Week 76: number analyzed (Participants) | 33
  Change from baseline T-score; Week 76 | -17.2 (15.71)
  Change from baseline T-score; Week 84: number analyzed (Participants) | 28
  Change from baseline T-score; Week 84 | -15.9 (13.93)
  Change from baseline T-score; Week 92: number analyzed (Participants) | 25
  Change from baseline T-score; Week 92 | -14.7 (16.41)
  Change from baseline T-score; Week 100: number analyzed (Participants) | 13
  Change from baseline T-score; Week 100 | -16.7 (17.47)
  Change from baseline T-score; Week 108: number analyzed (Participants) | 9
  Change from baseline T-score; Week 108 | -18.1 (20.59)
  Change from baseline T-score; Week 116: number analyzed (Participants) | 7
  Change from baseline T-score; Week 116 | -11.9 (18.25)
  Change from baseline T-score; Week 124: number analyzed (Participants) | 3
  Change from baseline T-score; Week 124 | -14.7 (27.30)

15. Secondary Outcome: Effect of SPN-812 on the "Inhibit" Scale in Adults With ADHD as Measured by the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A; Self Report)
Description: An additional secondary endpoint was the change from baseline in the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) "Inhibit" scale T-score by visit. The BRIEF-A is a 75-item self-rating scale that assesses overall functioning and 9 non-overlapping scales among 2 summary index scales. The "Inhibit" scale is one of four Behavioral Regulation Index-related scales; it captures the ability to control impulses and appropriately stop verbal, attentional, and physical behavior at the proper time. Subject's rate each item on a 3-point scale (1=Never, 2=Sometimes, or 3=Often) based on their experience in past month. The sum of 8 items yields the "Inhibit" raw score (range: 8-24), which is converted to a T-score (normative population mean=50 and standard deviation=10; T-score ≥ 65 is considered abnormally elevated). Post-baseline T-scores are converted to a change from baseline (CFB) T-score. A lower CFB "Inhibit" T-score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
T-score
  T-score; Baseline: number analyzed (Participants) | 157
  T-score; Baseline | 68.8 (9.83)
  Change from baseline T-score; Week 2: number analyzed (Participants) | 14
  Change from baseline T-score; Week 2 | -2.5 (10.16)
  Change from baseline T-score; Week 4: number analyzed (Participants) | 119
  Change from baseline T-score; Week 4 | -9.5 (9.57)
  Change from baseline T-score; Week 12: number analyzed (Participants) | 106
  Change from baseline T-score; Week 12 | -10.8 (10.90)
  Change from baseline T-score; Week 20: number analyzed (Participants) | 94
  Change from baseline T-score; Week 20 | -12.3 (11.54)
  Change from baseline T-score; Week 28: number analyzed (Participants) | 79
  Change from baseline T-score; Week 28 | -13.2 (11.27)
  Change from baseline T-score; Week 36: number analyzed (Participants) | 66
  Change from baseline T-score; Week 36 | -14.8 (11.13)
  Change from baseline T-score; Week 44: number analyzed (Participants) | 58
  Change from baseline T-score; Week 44 | -14.1 (10.59)
  Change from baseline T-score; Week 52: number analyzed (Participants) | 51
  Change from baseline T-score; Week 52 | -16.4 (12.93)
  Change from baseline T-score; Week 60: number analyzed (Participants) | 38
  Change from baseline T-score; Week 60 | -15.7 (12.10)
  Change from baseline T-score; Week 68: number analyzed (Participants) | 36
  Change from baseline T-score; Week 68 | -15.5 (12.07)
  Change from baseline T-score; Week 76: number analyzed (Participants) | 33
  Change from baseline T-score; Week 76 | -15.1 (13.24)
  Change from baseline T-score; Week 84: number analyzed (Participants) | 28
  Change from baseline T-score; Week 84 | -15.3 (9.49)
  Change from baseline T-score; Week 92: number analyzed (Participants) | 25
  Change from baseline T-score; Week 92 | -15.4 (11.94)
  Change from baseline T-score; Week 100: number analyzed (Participants) | 13
  Change from baseline T-score; Week 100 | -16.5 (12.19)
  Change from baseline T-score; Week 108: number analyzed (Participants) | 9
  Change from baseline T-score; Week 108 | -19.0 (15.88)
  Change from baseline T-score; Week 116: number analyzed (Participants) | 7
  Change from baseline T-score; Week 116 | -15.7 (12.72)
  Change from baseline T-score; Week 124: number analyzed (Participants) | 3
  Change from baseline T-score; Week 124 | -12.7 (22.03)

16. Secondary Outcome: Effect of SPN-812 on the "Self-Monitor" Scale in Adults With ADHD as Measured by the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A; Self Report)
Description: An additional secondary endpoint was the change from baseline in the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) "Self-Monitor" scale T-score by visit. The BRIEF-A is a 75-item self-rating scale that assesses overall functioning and 9 non-overlapping scales among 2 summary index scales. The "Self-Monitor" scale is one of four Behavioral Regulation Index-related scales; it reflects an individual's ability to recognize the effect of their own behavior on others. The subject rates each item on a 3-point scale (1=Never, 2=Sometimes, or 3=Often) based on their experience in past month. The sum of 6 items yields the "Self-Monitor" raw score (range: 6-18), which is converted to a T-score (normative population mean=50 and standard deviation=10; T-score ≥ 65 is considered abnormally elevated). Post-baseline T-scores are converted to a change from baseline (CFB) T-score. A lower CFB "Self-Monitor" T-score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
T-score
  T-score; Baseline: number analyzed (Participants) | 157
  T-score; Baseline | 60.4 (12.71)
  Change from baseline T-score; Week 2: number analyzed (Participants) | 14
  Change from baseline T-score; Week 2 | -0.7 (11.64)
  Change from baseline T-score; Week 4: number analyzed (Participants) | 119
  Change from baseline T-score; Week 4 | -7.8 (10.14)
  Change from baseline T-score; Week 12: number analyzed (Participants) | 106
  Change from baseline T-score; Week 12 | -7.2 (10.15)
  Change from baseline T-score; Week 20: number analyzed (Participants) | 94
  Change from baseline T-score; Week 20 | -9.5 (11.00)
  Change from baseline T-score; Week 28: number analyzed (Participants) | 79
  Change from baseline T-score; Week 28 | -10.3 (12.72)
  Change from baseline T-score; Week 36: number analyzed (Participants) | 66
  Change from baseline T-score; Week 36 | -11.3 (12.89)
  Change from baseline T-score; Week 44: number analyzed (Participants) | 58
  Change from baseline T-score; Week 44 | -10.9 (12.39)
  Change from baseline T-score; Week 52: number analyzed (Participants) | 51
  Change from baseline T-score; Week 52 | -11.3 (14.97)
  Change from baseline T-score; Week 60: number analyzed (Participants) | 38
  Change from baseline T-score; Week 60 | -10.1 (16.32)
  Change from baseline T-score; Week 68: number analyzed (Participants) | 36
  Change from baseline T-score; Week 68 | -11.6 (16.62)
  Change from baseline T-score; Week 76: number analyzed (Participants) | 33
  Change from baseline T-score; Week 76 | -11.3 (16.61)
  Change from baseline T-score; Week 84: number analyzed (Participants) | 28
  Change from baseline T-score; Week 84 | -9.9 (12.32)
  Change from baseline T-score; Week 92: number analyzed (Participants) | 25
  Change from baseline T-score; Week 92 | -9.0 (15.01)
  Change from baseline T-score; Week 100: number analyzed (Participants) | 13
  Change from baseline T-score; Week 100 | -7.5 (13.49)
  Change from baseline T-score; Week 108: number analyzed (Participants) | 9
  Change from baseline T-score; Week 108 | -6.6 (17.26)
  Change from baseline T-score; Week 116: number analyzed (Participants) | 7
  Change from baseline T-score; Week 116 | -2.9 (16.48)
  Change from baseline T-score; Week 124: number analyzed (Participants) | 3
  Change from baseline T-score; Week 124 | 1.0 (15.52)

17. Secondary Outcome: Effect of SPN-812 on the "Plan/Organize" Scale in Adults With ADHD as Measured by the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A; Self Report)
Description: An additional secondary endpoint was the change from baseline in the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) "Plan/Organize" scale T-score by visit. The BRIEF-A is a 75-item self-rating scale that assesses overall functioning and 9 non-overlapping scales among 2 summary index scales. The "Plan/Organize" scale is one of five Metacognition Index-related scales; captures an individual's ability to anticipate events, set goals, pre-plan, organize, and carry out tasks systematically. Subjects rate each item on a 3-point scale (1=Never, 2=Sometimes, 3=Often) based on their experience in past month. The sum of 10 items yields the "Plan/Organize" raw score (range: 10-30), which is converted to a T-score (normative population mean=50 and standard deviation=10; T-score ≥65 is considered abnormally elevated). Post-baseline T-scores are converted to a change from baseline (CFB) T-score. A lower CFB "Plan/Organize" T-score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
T-score
  T-score; Baseline: number analyzed (Participants) | 157
  T-score; Baseline | 70.6 (12.62)
  Change from baseline T-score; Week 2: number analyzed (Participants) | 14
  Change from baseline T-score; Week 2 | 0.1 (11.71)
  Change from baseline T-score; Week 4: number analyzed (Participants) | 119
  Change from baseline T-score; Week 4 | -8.5 (10.94)
  Change from baseline T-score; Week 12: number analyzed (Participants) | 106
  Change from baseline T-score; Week 12 | -8.6 (11.87)
  Change from baseline T-score; Week 20: number analyzed (Participants) | 93
  Change from baseline T-score; Week 20 | -12.0 (13.29)
  Change from baseline T-score; Week 28: number analyzed (Participants) | 79
  Change from baseline T-score; Week 28 | -13.2 (13.20)
  Change from baseline T-score; Week 36: number analyzed (Participants) | 66
  Change from baseline T-score; Week 36 | -13.2 (12.47)
  Change from baseline T-score; Week 44: number analyzed (Participants) | 58
  Change from baseline T-score; Week 44 | -12.1 (12.21)
  Change from baseline T-score; Week 52: number analyzed (Participants) | 51
  Change from baseline T-score; Week 52 | -12.7 (12.49)
  Change from baseline T-score; Week 60: number analyzed (Participants) | 38
  Change from baseline T-score; Week 60 | -13.7 (13.28)
  Change from baseline T-score; Week 68: number analyzed (Participants) | 36
  Change from baseline T-score; Week 68 | -14.3 (15.35)
  Change from baseline T-score; Week 76: number analyzed (Participants) | 33
  Change from baseline T-score; Week 76 | -14.4 (14.32)
  Change from baseline T-score; Week 84: number analyzed (Participants) | 28
  Change from baseline T-score; Week 84 | -13.3 (14.49)
  Change from baseline T-score; Week 92: number analyzed (Participants) | 25
  Change from baseline T-score; Week 92 | -12.8 (17.07)
  Change from baseline T-score; Week 100: number analyzed (Participants) | 13
  Change from baseline T-score; Week 100 | -14.2 (18.32)
  Change from baseline T-score; Week 108: number analyzed (Participants) | 9
  Change from baseline T-score; Week 108 | -15.3 (19.50)
  Change from baseline T-score; Week 116: number analyzed (Participants) | 7
  Change from baseline T-score; Week 116 | -11.7 (16.73)
  Change from baseline T-score; Week 124: number analyzed (Participants) | 3
  Change from baseline T-score; Week 124 | -17.3 (25.32)

18. Secondary Outcome: Effect of SPN-812 on the "Shift" Scale in Adults With ADHD as Measured by the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A; Self Report)
Description: An additional secondary endpoint was the change from baseline in the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) "Shift" scale T-score by visit. The BRIEF-A is a 75-item self-rating scale that assesses overall functioning and 9 non-overlapping scales among 2 summary index scales. The "Shift" scale is one of four Behavioral Regulation Index-related scales; it captures one's ability to move freely from one situation/activity/aspect of a problem to another and think flexibly to aid problem-solving. Subjects rate each item on a 3-point scale (1=Never, 2=Sometimes, or 3=Often) based on their experience in past month. The sum of 6 items yields the "Shift" raw score (range: 6-18), which is converted to a T-score (normative population mean=50 and standard deviation=10; T-score ≥ 65 is considered abnormally elevated). Post-baseline T-scores are converted to a change from baseline (CFB) T-score. A lower CFB "Shift" T-score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
T-score
  T-score; Baseline: number analyzed (Participants) | 157
  T-score; Baseline | 63.7 (12.34)
  Change from baseline T-score; Week 2: number analyzed (Participants) | 14
  Change from baseline T-score; Week 2 | -1.9 (9.41)
  Change from baseline T-score; Week 4: number analyzed (Participants) | 119
  Change from baseline T-score; Week 4 | -7.3 (10.65)
  Change from baseline T-score; Week 12: number analyzed (Participants) | 106
  Change from baseline T-score; Week 12 | -8.2 (12.22)
  Change from baseline T-score; Week 20: number analyzed (Participants) | 94
  Change from baseline T-score; Week 20 | -8.9 (13.26)
  Change from baseline T-score; Week 28: number analyzed (Participants) | 79
  Change from baseline T-score; Week 28 | -9.4 (12.54)
  Change from baseline T-score; Week 36: number analyzed (Participants) | 66
  Change from baseline T-score; Week 36 | -9.7 (11.30)
  Change from baseline T-score; Week 44: number analyzed (Participants) | 58
  Change from baseline T-score; Week 44 | -8.6 (12.31)
  Change from baseline T-score; Week 52: number analyzed (Participants) | 51
  Change from baseline T-score; Week 52 | -9.0 (13.40)
  Change from baseline T-score; Week 60: number analyzed (Participants) | 38
  Change from baseline T-score; Week 60 | -8.5 (13.23)
  Change from baseline T-score; Week 68: number analyzed (Participants) | 36
  Change from baseline T-score; Week 68 | -9.6 (14.08)
  Change from baseline T-score; Week 76: number analyzed (Participants) | 33
  Change from baseline T-score; Week 76 | -10.7 (12.35)
  Change from baseline T-score; Week 84: number analyzed (Participants) | 28
  Change from baseline T-score; Week 84 | -10.4 (11.63)
  Change from baseline T-score; Week 92: number analyzed (Participants) | 25
  Change from baseline T-score; Week 92 | -9.1 (12.37)
  Change from baseline T-score; Week 100: number analyzed (Participants) | 13
  Change from baseline T-score; Week 100 | -11.5 (12.43)
  Change from baseline T-score; Week 108: number analyzed (Participants) | 9
  Change from baseline T-score; Week 108 | -13.7 (17.28)
  Change from baseline T-score; Week 116: number analyzed (Participants) | 7
  Change from baseline T-score; Week 116 | -12.1 (14.88)
  Change from baseline T-score; Week 124: number analyzed (Participants) | 3
  Change from baseline T-score; Week 124 | -13.7 (30.60)

19. Secondary Outcome: Effect of SPN-812 on the "Initiate" Scale in Adults With ADHD as Measured by the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A; Self Report)
Description: An additional secondary endpoint was the change from baseline in the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) "Initiate" scale T-score by visit. The BRIEF-A is a 75-item self-rating scale that assesses overall functioning and 9 non-overlapping scales among 2 summary index scales. The "Initiate" scale is one of five Metacognition Index-related scales; it captures an individual's ability to begin a task or activity without external prompting and to independently generate ideas. Subjects rate each item on a 3-point scale (1=Never, 2=Sometimes, or 3=Often) based on their experience in past month. The sum of 8 items yields the "Initiate" scale raw score (range: 8-24), which is converted to a T-score (normative population mean=50 and standard deviation=10; T-score ≥ 65 is considered abnormally elevated). Post-baseline T-scores are converted to a change from baseline (CFB) T-score. A lower CFB "Initiate" T-score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
T-score
  T-score; Baseline: number analyzed (Participants) | 156
  T-score; Baseline | 68.0 (10.83)
  Change from baseline T-score; Week 2: number analyzed (Participants) | 14
  Change from baseline T-score; Week 2 | 1.9 (8.59)
  Change from baseline T-score; Week 4: number analyzed (Participants) | 118
  Change from baseline T-score; Week 4 | -6.2 (10.68)
  Change from baseline T-score; Week 12: number analyzed (Participants) | 105
  Change from baseline T-score; Week 12 | -8.0 (12.01)
  Change from baseline T-score; Week 20: number analyzed (Participants) | 93
  Change from baseline T-score; Week 20 | -9.8 (12.96)
  Change from baseline T-score; Week 28: number analyzed (Participants) | 78
  Change from baseline T-score; Week 28 | -11.7 (12.53)
  Change from baseline T-score; Week 36: number analyzed (Participants) | 65
  Change from baseline T-score; Week 36 | -11.6 (11.89)
  Change from baseline T-score; Week 44: number analyzed (Participants) | 57
  Change from baseline T-score; Week 44 | -10.7 (11.25)
  Change from baseline T-score; Week 52: number analyzed (Participants) | 50
  Change from baseline T-score; Week 52 | -11.7 (13.64)
  Change from baseline T-score; Week 60: number analyzed (Participants) | 38
  Change from baseline T-score; Week 60 | -12.1 (13.16)
  Change from baseline T-score; Week 68: number analyzed (Participants) | 36
  Change from baseline T-score; Week 68 | -14.4 (13.61)
  Change from baseline T-score; Week 76: number analyzed (Participants) | 33
  Change from baseline T-score; Week 76 | -15.9 (13.81)
  Change from baseline T-score; Week 84: number analyzed (Participants) | 28
  Change from baseline T-score; Week 84 | -12.7 (11.31)
  Change from baseline T-score; Week 92: number analyzed (Participants) | 25
  Change from baseline T-score; Week 92 | -12.0 (13.09)
  Change from baseline T-score; Week 100: number analyzed (Participants) | 13
  Change from baseline T-score; Week 100 | -15.0 (13.23)
  Change from baseline T-score; Week 108: number analyzed (Participants) | 9
  Change from baseline T-score; Week 108 | -14.0 (14.21)
  Change from baseline T-score; Week 116: number analyzed (Participants) | 7
  Change from baseline T-score; Week 116 | -11.9 (10.76)
  Change from baseline T-score; Week 124: number analyzed (Participants) | 3
  Change from baseline T-score; Week 124 | -13.7 (18.48)

20. Secondary Outcome: Effect of SPN-812 on the "Task Monitor" Scale in Adults With ADHD as Measured by the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A; Self Report)
Description: An additional secondary endpoint was the change from baseline in the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) "Task Monitor" scale T-score by visit. The BRIEF-A is a 75-item self-rating scale that assesses overall functioning and 9 non-overlapping scales among 2 summary index scales. The "Task Monitor" scale is one of five Metacognition Index-related scales; it captures an individual's ability to assess performance for mistakes during or after finishing a task. The subject rates each item on a 3-point scale (1=Never, 2=Sometimes, or 3=Often) based on their experience in past month. The sum of 6 items yields the "Task Monitor" raw score (range: 6-18), which is converted to a T-score (normative population mean=50 and standard deviation=10; T-score ≥ 65 is considered abnormally elevated). Post-baseline T-scores are converted to a change from baseline (CFB) T-score. A lower CFB "Task Monitor" T-score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
T-score
  T-score; Baseline: number analyzed (Participants) | 157
  T-score; Baseline | 71.1 (11.67)
  Change from baseline T-score; Week 2: number analyzed (Participants) | 14
  Change from baseline T-score; Week 2 | -1.4 (9.46)
  Change from baseline T-score; Week 4: number analyzed (Participants) | 119
  Change from baseline T-score; Week 4 | -7.6 (11.14)
  Change from baseline T-score; Week 12: number analyzed (Participants) | 105
  Change from baseline T-score; Week 12 | -8.4 (11.70)
  Change from baseline T-score; Week 20: number analyzed (Participants) | 94
  Change from baseline T-score; Week 20 | -10.2 (13.68)
  Change from baseline T-score; Week 28: number analyzed (Participants) | 79
  Change from baseline T-score; Week 28 | -13.0 (12.57)
  Change from baseline T-score; Week 36: number analyzed (Participants) | 66
  Change from baseline T-score; Week 36 | -12.7 (12.79)
  Change from baseline T-score; Week 44: number analyzed (Participants) | 58
  Change from baseline T-score; Week 44 | -12.8 (12.33)
  Change from baseline T-score; Week 52: number analyzed (Participants) | 51
  Change from baseline T-score; Week 52 | -14.1 (14.99)
  Change from baseline T-score; Week 60: number analyzed (Participants) | 38
  Change from baseline T-score; Week 60 | -16.4 (15.23)
  Change from baseline T-score; Week 68: number analyzed (Participants) | 36
  Change from baseline T-score; Week 68 | -14.9 (16.02)
  Change from baseline T-score; Week 76: number analyzed (Participants) | 33
  Change from baseline T-score; Week 76 | -16.1 (15.82)
  Change from baseline T-score; Week 84: number analyzed (Participants) | 28
  Change from baseline T-score; Week 84 | -13.4 (16.15)
  Change from baseline T-score; Week 92: number analyzed (Participants) | 25
  Change from baseline T-score; Week 92 | -11.3 (19.47)
  Change from baseline T-score; Week 100: number analyzed (Participants) | 13
  Change from baseline T-score; Week 100 | -14.1 (19.74)
  Change from baseline T-score; Week 108: number analyzed (Participants) | 9
  Change from baseline T-score; Week 108 | -14.7 (21.50)
  Change from baseline T-score; Week 116: number analyzed (Participants) | 7
  Change from baseline T-score; Week 116 | -7.9 (22.39)
  Change from baseline T-score; Week 124: number analyzed (Participants) | 3
  Change from baseline T-score; Week 124 | -9.3 (21.83)

21. Secondary Outcome: Effect of SPN-812 on the "Emotional Control" Scale in Adults With ADHD as Measured by the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A; Self Report)
Description: An additional secondary endpoint was the change from baseline in the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) "Emotional Control" scale T-score by visit. The BRIEF-A is a 75-item self-rating scale that assesses overall functioning and 9 non-overlapping scales among 2 summary index scales. The "Emotional Control" scale is one of four Behavioral Regulation Index-related scales; it captures an individual's ability to modulate their emotional responses appropriately. Subjects rate each item on a 3-point scale (1=Never, 2=Sometimes, or 3=Often) based on their experience in past month. The sum of 10 items yields the "Emotional Control" raw score (range: 10-30), which is converted to a T-score (normative population mean=50 and standard deviation=10; T-score ≥ 65 is considered abnormally elevated). Post-baseline T-scores are converted to a change from baseline (CFB) T-score. A lower CFB "Emotional Control" T-score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
T-score
  T-score; Baseline: number analyzed (Participants) | 157
  T-score; Baseline | 53.5 (11.95)
  Change from baseline T-score; Week 2: number analyzed (Participants) | 14
  Change from baseline T-score; Week 2 | 1.5 (5.27)
  Change from baseline T-score; Week 4: number analyzed (Participants) | 119
  Change from baseline T-score; Week 4 | -4.5 (9.38)
  Change from baseline T-score; Week 12: number analyzed (Participants) | 106
  Change from baseline T-score; Week 12 | -4.0 (10.35)
  Change from baseline T-score; Week 20: number analyzed (Participants) | 94
  Change from baseline T-score; Week 20 | -5.6 (9.90)
  Change from baseline T-score; Week 28: number analyzed (Participants) | 79
  Change from baseline T-score; Week 28 | -4.7 (11.22)
  Change from baseline T-score; Week 36: number analyzed (Participants) | 66
  Change from baseline T-score; Week 36 | -5.1 (10.36)
  Change from baseline T-score; Week 44: number analyzed (Participants) | 58
  Change from baseline T-score; Week 44 | -4.5 (9.74)
  Change from baseline T-score; Week 52: number analyzed (Participants) | 51
  Change from baseline T-score; Week 52 | -5.5 (11.38)
  Change from baseline T-score; Week 60: number analyzed (Participants) | 38
  Change from baseline T-score; Week 60 | -5.5 (11.30)
  Change from baseline T-score; Week 68: number analyzed (Participants) | 36
  Change from baseline T-score; Week 68 | -6.6 (13.00)
  Change from baseline T-score; Week 76: number analyzed (Participants) | 33
  Change from baseline T-score; Week 76 | -7.4 (11.97)
  Change from baseline T-score; Week 84: number analyzed (Participants) | 28
  Change from baseline T-score; Week 84 | -8.1 (11.72)
  Change from baseline T-score; Week 92: number analyzed (Participants) | 25
  Change from baseline T-score; Week 92 | -7.0 (10.51)
  Change from baseline T-score; Week 100: number analyzed (Participants) | 13
  Change from baseline T-score; Week 100 | -7.6 (11.23)
  Change from baseline T-score; Week 108: number analyzed (Participants) | 9
  Change from baseline T-score; Week 108 | -9.8 (16.01)
  Change from baseline T-score; Week 116: number analyzed (Participants) | 7
  Change from baseline T-score; Week 116 | -10.4 (12.79)
  Change from baseline T-score; Week 124: number analyzed (Participants) | 3
  Change from baseline T-score; Week 124 | -6.7 (16.50)

22. Secondary Outcome: Effect of SPN-812 on the "Working Memory" Scale in Adults With ADHD as Measured by the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A; Self Report)
Description: An additional secondary endpoint was the change from baseline in the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) "Working Memory" scale T-score by visit. The BRIEF-A is a 75-item self-rating scale that assesses overall functioning and 9 non-overlapping scales among 2 summary index scales. The "Working Memory" scale is one of five Metacognition Index-related scales; it captures one's ability to hold information in mind in order to complete a task and stay with, or stick to, an activity. Subjects rate each item on a 3-point scale (1=Never, 2=Sometimes, 3=Often) based on their experience in past month. The sum of 8 items yields the "Working Memory" raw score (range: 8-24), which is converted to a T-score (normative population mean=50 and standard deviation=10; T-score ≥65 is considered abnormally elevated). Post-baseline T-scores are converted to a change from baseline (CFB) T-score. A lower CFB "Working Memory" T-score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
T-score
  T-score; Baseline: number analyzed (Participants) | 157
  T-score; Baseline | 77.4 (10.59)
  Change from baseline T-score; Week 2: number analyzed (Participants) | 14
  Change from baseline T-score; Week 2 | -6.2 (11.29)
  Change from baseline T-score; Week 4: number analyzed (Participants) | 118
  Change from baseline T-score; Week 4 | -9.7 (11.22)
  Change from baseline T-score; Week 12: number analyzed (Participants) | 106
  Change from baseline T-score; Week 12 | -11.8 (12.73)
  Change from baseline T-score; Week 20: number analyzed (Participants) | 94
  Change from baseline T-score; Week 20 | -14.0 (13.12)
  Change from baseline T-score; Week 28: number analyzed (Participants) | 79
  Change from baseline T-score; Week 28 | -15.5 (13.44)
  Change from baseline T-score; Week 36: number analyzed (Participants) | 66
  Change from baseline T-score; Week 36 | -15.6 (12.70)
  Change from baseline T-score; Week 44: number analyzed (Participants) | 58
  Change from baseline T-score; Week 44 | -17.2 (11.91)
  Change from baseline T-score; Week 52: number analyzed (Participants) | 51
  Change from baseline T-score; Week 52 | -16.8 (14.43)
  Change from baseline T-score; Week 60: number analyzed (Participants) | 38
  Change from baseline T-score; Week 60 | -17.0 (14.74)
  Change from baseline T-score; Week 68: number analyzed (Participants) | 36
  Change from baseline T-score; Week 68 | -16.9 (15.92)
  Change from baseline T-score; Week 76: number analyzed (Participants) | 33
  Change from baseline T-score; Week 76 | -17.0 (15.57)
  Change from baseline T-score; Week 84: number analyzed (Participants) | 28
  Change from baseline T-score; Week 84 | -18.4 (13.12)
  Change from baseline T-score; Week 92: number analyzed (Participants) | 25
  Change from baseline T-score; Week 92 | -17.4 (14.56)
  Change from baseline T-score; Week 100: number analyzed (Participants) | 13
  Change from baseline T-score; Week 100 | -15.2 (18.48)
  Change from baseline T-score; Week 108: number analyzed (Participants) | 9
  Change from baseline T-score; Week 108 | -18.2 (20.52)
  Change from baseline T-score; Week 116: number analyzed (Participants) | 7
  Change from baseline T-score; Week 116 | -7.0 (18.65)
  Change from baseline T-score; Week 124: number analyzed (Participants) | 3
  Change from baseline T-score; Week 124 | -11.0 (27.22)

23. Secondary Outcome: Effect of SPN-812 on "Organization of Materials" Scale in Adults With ADHD as Measured by the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A; Self Report)
Description: An additional secondary endpoint was the change from baseline in the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) "Organization of Materials" scale T-score by visit. The BRIEF-A is a 75-item self-rating scale that assesses overall functioning and 9 non-overlapping scales among 2 summary index scales. The "Organization of Materials" scale is one of five Metacognition Index-related scales; it captures one's ability to keep areas orderly and maintain materials. Subjects rate each item on a 3-point scale (1=Never, 2=Sometimes, 3=Often) based on their experience in past month. The sum of 8 items yields the "Organization of Materials" raw score (range: 8-24), which is converted to a T-score (normative population mean=50 and standard deviation=10; T-score ≥ 65 is considered abnormally elevated). Post-baseline T-scores are converted to a change from baseline (CFB) T-score. A lower CFB "Organization of Materials" T-score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
T-score
  T-score; Baseline: number analyzed (Participants) | 157
  T-score; Baseline | 64.4 (12.22)
  Change from baseline T-score; Week 2: number analyzed (Participants) | 14
  Change from baseline T-score; Week 2 | -5.3 (9.88)
  Change from baseline T-score; Week 4: number analyzed (Participants) | 119
  Change from baseline T-score; Week 4 | -6.9 (9.11)
  Change from baseline T-score; Week 12: number analyzed (Participants) | 105
  Change from baseline T-score; Week 12 | -7.8 (10.25)
  Change from baseline T-score; Week 20: number analyzed (Participants) | 93
  Change from baseline T-score; Week 20 | -8.7 (11.51)
  Change from baseline T-score; Week 28: number analyzed (Participants) | 79
  Change from baseline T-score; Week 28 | -11.1 (10.77)
  Change from baseline T-score; Week 36: number analyzed (Participants) | 66
  Change from baseline T-score; Week 36 | -11.7 (11.23)
  Change from baseline T-score; Week 44: number analyzed (Participants) | 58
  Change from baseline T-score; Week 44 | -11.3 (11.25)
  Change from baseline T-score; Week 52: number analyzed (Participants) | 51
  Change from baseline T-score; Week 52 | -11.2 (11.33)
  Change from baseline T-score; Week 60: number analyzed (Participants) | 38
  Change from baseline T-score; Week 60 | -11.8 (11.95)
  Change from baseline T-score; Week 68: number analyzed (Participants) | 36
  Change from baseline T-score; Week 68 | -12.5 (12.29)
  Change from baseline T-score; Week 76: number analyzed (Participants) | 33
  Change from baseline T-score; Week 76 | -11.5 (13.34)
  Change from baseline T-score; Week 84: number analyzed (Participants) | 28
  Change from baseline T-score; Week 84 | -10.4 (12.45)
  Change from baseline T-score; Week 92: number analyzed (Participants) | 25
  Change from baseline T-score; Week 92 | -10.4 (12.47)
  Change from baseline T-score; Week 100: number analyzed (Participants) | 13
  Change from baseline T-score; Week 100 | -12.5 (13.94)
  Change from baseline T-score; Week 108: number analyzed (Participants) | 9
  Change from baseline T-score; Week 108 | -14.4 (17.88)
  Change from baseline T-score; Week 116: number analyzed (Participants) | 7
  Change from baseline T-score; Week 116 | -10.3 (15.52)
  Change from baseline T-score; Week 124: number analyzed (Participants) | 3
  Change from baseline T-score; Week 124 | -10.3 (26.08)

24. Secondary Outcome: Effect of SPN-812 on Overall Symptoms of Depression in Adults With ADHD as Measured by the Symptoms of Depression Questionnaire (SDQ)
Description: An additional secondary endpoint was the change from baseline in the Symptoms of Depression Questionnaire (SDQ) Total Score by visit. The SDQ is a 44-item self-rating scale assessing overall depression and 5 related symptoms/subscales, including items related to lassitude, mood, and cognitive functioning (18 items; SDQ-1); anxiety, agitation, irritability, and anger (13 items; SDQ-2); suicidal ideation (6 items; SDQ-3); disruptions in sleep quality (3 items; SDQ-4); and changes in appetite and weight (4 items; SDQ-5). Each item is rated on a 6-point scale based on a subject's perception in past month of what is normal (score = 2), what is better than normal (score = 1), and what is worse than normal (scores = 3-6). The sum of 44 items yields the raw Total score (range: 44-264); a higher Total score indicates worse depression. Post-baseline raw Total scores are converted to a change from baseline score. A lower change from baseline Total score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: Safety Population (N), defined as subjects who signed Informed Consent and took at least 1 dose of SPN-812. At each Visit/Week, data is summarized with descriptive statistics for the number of subjects analyzed (n; subjects with a valid SDQ assessment at baseline [pre-dosing] and at the respective post-baseline [after first dose] Visit/Week). Due to attrition and/or missing data, the number of subjects analyzed at each Visit/Week may be less than and unequal to Safety Population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
units on a scale
  Raw score; Baseline: number analyzed (Participants) | 158
  Raw score; Baseline | 105.9 (17.18)
  Change from baseline score; Week 2: number analyzed (Participants) | 14
  Change from baseline score; Week 2 | 4.8 (17.03)
  Change from baseline score; Week 4: number analyzed (Participants) | 121
  Change from baseline score; Week 4 | -2.7 (14.57)
  Change from baseline score; Week 12: number analyzed (Participants) | 109
  Change from baseline score; Week 12 | -1.9 (19.79)
  Change from baseline score; Week 20: number analyzed (Participants) | 94
  Change from baseline score; Week 20 | -3.8 (16.50)
  Change from baseline score; Week 28: number analyzed (Participants) | 79
  Change from baseline score; Week 28 | -3.5 (17.24)
  Change from baseline score; Week 36: number analyzed (Participants) | 67
  Change from baseline score; Week 36 | -2.7 (17.15)
  Change from baseline score; Week 44: number analyzed (Participants) | 59
  Change from baseline score; Week 44 | -6.2 (16.56)
  Change from baseline score; Week 52: number analyzed (Participants) | 51
  Change from baseline score; Week 52 | -4.0 (19.22)
  Change from baseline score; Week 60: number analyzed (Participants) | 38
  Change from baseline score; Week 60 | -5.3 (15.63)
  Change from baseline score; Week 68: number analyzed (Participants) | 35
  Change from baseline score; Week 68 | -5.9 (20.64)
  Change from baseline score; Week 76: number analyzed (Participants) | 33
  Change from baseline score; Week 76 | -8.2 (15.11)
  Change from baseline score; Week 84: number analyzed (Participants) | 29
  Change from baseline score; Week 84 | -7.1 (12.49)
  Change from baseline score; Week 92: number analyzed (Participants) | 25
  Change from baseline score; Week 92 | -8.4 (12.83)
  Change from baseline score; Week 100: number analyzed (Participants) | 13
  Change from baseline score; Week 100 | -6.4 (11.61)
  Change from baseline score; Week 108: number analyzed (Participants) | 9
  Change from baseline score; Week 108 | -2.9 (20.37)
  Change from baseline score; Week 116: number analyzed (Participants) | 7
  Change from baseline score; Week 116 | -3.6 (18.19)
  Change from baseline score; Week 124: number analyzed (Participants) | 4
  Change from baseline score; Week 124 | -9.0 (13.74)

25. Secondary Outcome: Effect of SPN-812 on "Lassitude, Mood, and Cognitive Functioning" (SDQ-1) Subscale in Adults With ADHD as Measured by the Symptoms of Depression Questionnaire (SDQ)
Description: An additional secondary endpoint was the change from baseline in the Symptoms of Depression Questionnaire (SDQ) "Lassitude, Mood, and Cognitive Functioning" (SDQ-1) Subscale Score by visit. The SDQ is a 44-item self-rating scale assessing overall depression and 5 related symptoms/subscales, including 18 items related to lassitude, mood, and cognitive functioning (SDQ-1 subscale). Each item is rated on a 6-point scale based on a subject's perception in past month of what is normal (score = 2), what is better than normal (score = 1), and what is worse than normal (scores = 3-6). The sum of these 18 items yields the raw SDQ-1 subscale score (range: 17-102); a higher SDQ-1 subscale score indicates worse lassitude, mood, and cognitive functioning. Post-baseline raw SDQ-1 subscale scores are converted to a change from baseline score. A lower change from baseline SDQ-1 subscale score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
units on a scale
  Raw score; Baseline: number analyzed (Participants) | 158
  Raw score; Baseline | 45.6 (9.40)
  Change from baseline score; Week 2: number analyzed (Participants) | 14
  Change from baseline score; Week 2 | 0.5 (9.55)
  Change from baseline score; Week 4: number analyzed (Participants) | 121
  Change from baseline score; Week 4 | -2.4 (7.94)
  Change from baseline score; Week 12: number analyzed (Participants) | 109
  Change from baseline score; Week 12 | -2.3 (10.70)
  Change from baseline score; Week 20: number analyzed (Participants) | 95
  Change from baseline score; Week 20 | -3.0 (9.95)
  Change from baseline score; Week 28: number analyzed (Participants) | 80
  Change from baseline score; Week 28 | -3.2 (10.28)
  Change from baseline score; Week 36: number analyzed (Participants) | 67
  Change from baseline score; Week 36 | -2.7 (9.99)
  Change from baseline score; Week 44: number analyzed (Participants) | 59
  Change from baseline score; Week 44 | -4.0 (10.14)
  Change from baseline score; Week 52: number analyzed (Participants) | 51
  Change from baseline score; Week 52 | -3.3 (11.01)
  Change from baseline score; Week 60: number analyzed (Participants) | 38
  Change from baseline score; Week 60 | -4.2 (10.64)
  Change from baseline score; Week 68: number analyzed (Participants) | 35
  Change from baseline score; Week 68 | -3.9 (12.79)
  Change from baseline score; Week 76: number analyzed (Participants) | 33
  Change from baseline score; Week 76 | -5.4 (10.31)
  Change from baseline score; Week 84: number analyzed (Participants) | 29
  Change from baseline score; Week 84 | -3.9 (6.46)
  Change from baseline score; Week 92: number analyzed (Participants) | 25
  Change from baseline score; Week 92 | -3.8 (7.74)
  Change from baseline score; Week 100: number analyzed (Participants) | 13
  Change from baseline score; Week 100 | -2.6 (6.37)
  Change from baseline score; Week 108: number analyzed (Participants) | 9
  Change from baseline score; Week 108 | -2.1 (9.55)
  Change from baseline score; Week 116: number analyzed (Participants) | 7
  Change from baseline score; Week 116 | -1.7 (8.50)
  Change from baseline score; Week 124: number analyzed (Participants) | 4
  Change from baseline score; Week 124 | -5.8 (8.02)

26. Secondary Outcome: Effect of SPN-812 on "Anxiety, Agitation, Irritability, and Anger" (SDQ-2) Subscale in Adults With ADHD as Measured by the Symptoms of Depression Questionnaire (SDQ)
Description: An additional secondary endpoint was the change from baseline in the Symptoms of Depression Questionnaire (SDQ) "Anxiety, Agitation, Irritability, and Anger" (SDQ-2) Score by visit. The SDQ is a 44-item self-rating scale assessing overall depression and 5 related symptoms/subscales, including 13 items related to anxiety, agitation, irritability, and anger (SDQ-2 subscale). Each item is rated on a 6-point scale based on a subject's perception in past month of what is normal (score = 2), what is better than normal (score = 1), and what is worse than normal (scores = 3-6). The sum of these 13 items yields the raw SDQ-2 subscale score (range: 13-78); a higher SDQ-2 subscale score indicates worse anxiety, agitation, irritability, and anger. Post-baseline raw SDQ-2 subscale scores are converted to a change from baseline score. A lower change from baseline SDQ-2 subscale score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
units on a scale
  Raw score; Baseline: number analyzed (Participants) | 158
  Raw score; Baseline | 31.1 (5.93)
  Change from baseline score; Week 2: number analyzed (Participants) | 14
  Change from baseline score; Week 2 | 2.6 (4.86)
  Change from baseline score; Week 4: number analyzed (Participants) | 121
  Change from baseline score; Week 4 | -0.6 (5.49)
  Change from baseline score; Week 12: number analyzed (Participants) | 109
  Change from baseline score; Week 12 | 0.0 (6.97)
  Change from baseline score; Week 20: number analyzed (Participants) | 95
  Change from baseline score; Week 20 | -0.6 (5.70)
  Change from baseline score; Week 28: number analyzed (Participants) | 80
  Change from baseline score; Week 28 | -0.6 (5.79)
  Change from baseline score; Week 36: number analyzed (Participants) | 67
  Change from baseline score; Week 36 | 0.0 (6.07)
  Change from baseline score; Week 44: number analyzed (Participants) | 59
  Change from baseline score; Week 44 | -1.4 (5.18)
  Change from baseline score; Week 52: number analyzed (Participants) | 51
  Change from baseline score; Week 52 | -0.7 (5.23)
  Change from baseline score; Week 60: number analyzed (Participants) | 38
  Change from baseline score; Week 60 | -0.9 (4.66)
  Change from baseline score; Week 68: number analyzed (Participants) | 35
  Change from baseline score; Week 68 | -0.8 (5.96)
  Change from baseline score; Week 76: number analyzed (Participants) | 33
  Change from baseline score; Week 76 | -1.8 (4.32)
  Change from baseline score; Week 84: number analyzed (Participants) | 29
  Change from baseline score; Week 84 | -1.2 (4.87)
  Change from baseline score; Week 92: number analyzed (Participants) | 25
  Change from baseline score; Week 92 | -2.9 (4.59)
  Change from baseline score; Week 100: number analyzed (Participants) | 13
  Change from baseline score; Week 100 | -2.3 (3.88)
  Change from baseline score; Week 108: number analyzed (Participants) | 9
  Change from baseline score; Week 108 | 0.1 (6.62)
  Change from baseline score; Week 116: number analyzed (Participants) | 7
  Change from baseline score; Week 116 | -0.4 (5.29)
  Change from baseline score; Week 124: number analyzed (Participants) | 4
  Change from baseline score; Week 124 | -1.0 (4.55)

27. Secondary Outcome: Effect of SPN-812 on "Suicidal Ideation" (SDQ-3) Subscale in Adults With ADHD as Measured by the Symptoms of Depression Questionnaire (SDQ)
Description: An additional secondary endpoint was the change from baseline in the Symptoms of Depression Questionnaire (SDQ) "Suicidal Ideation" (SDQ-3) Subscale by visit. The SDQ is a 44-item self-rating scale assessing overall depression and 5 related symptoms/subscales, including 6 items related to suicidal ideation (SDQ-3). Each item is rated on a 6-point scale based on a subject's perception in past month of what is normal (score = 2), what is better than normal (score = 1), and what is worse than normal (scores = 3-6). The sum of these 6 items yields the raw SDQ-3 subscale score (range: 6-36); a higher SDQ-3 subscale score indicates worse "suicidal ideation". Post-baseline raw SDQ-3 subscale scores are converted to a change from baseline score. A lower change from baseline SDQ-3 subscale score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
units on a scale
  Raw score; Baseline: number analyzed (Participants) | 158
  Raw score; Baseline | 12.4 (1.92)
  Change from baseline score; Week 2: number analyzed (Participants) | 14
  Change from baseline score; Week 2 | 0.3 (2.61)
  Change from baseline score; Week 4: number analyzed (Participants) | 121
  Change from baseline score; Week 4 | -0.1 (2.06)
  Change from baseline score; Week 12: number analyzed (Participants) | 109
  Change from baseline score; Week 12 | -0.1 (2.53)
  Change from baseline score; Week 20: number analyzed (Participants) | 95
  Change from baseline score; Week 20 | 0.0 (2.31)
  Change from baseline score; Week 28: number analyzed (Participants) | 80
  Change from baseline score; Week 28 | 0.1 (2.08)
  Change from baseline score; Week 36: number analyzed (Participants) | 67
  Change from baseline score; Week 36 | 0.3 (2.63)
  Change from baseline score; Week 44: number analyzed (Participants) | 59
  Change from baseline score; Week 44 | -0.1 (2.13)
  Change from baseline score; Week 52: number analyzed (Participants) | 51
  Change from baseline score; Week 52 | 0.4 (2.80)
  Change from baseline score; Week 60: number analyzed (Participants) | 38
  Change from baseline score; Week 60 | 0.0 (1.99)
  Change from baseline score; Week 68: number analyzed (Participants) | 35
  Change from baseline score; Week 68 | -0.2 (2.19)
  Change from baseline score; Week 76: number analyzed (Participants) | 33
  Change from baseline score; Week 76 | -0.3 (1.90)
  Change from baseline score; Week 84: number analyzed (Participants) | 29
  Change from baseline score; Week 84 | -0.3 (1.79)
  Change from baseline score; Week 92: number analyzed (Participants) | 25
  Change from baseline score; Week 92 | -0.5 (1.39)
  Change from baseline score; Week 100: number analyzed (Participants) | 13
  Change from baseline score; Week 100 | -0.8 (1.42)
  Change from baseline score; Week 108: number analyzed (Participants) | 9
  Change from baseline score; Week 108 | 0.3 (1.73)
  Change from baseline score; Week 116: number analyzed (Participants) | 7
  Change from baseline score; Week 116 | -0.3 (1.89)
  Change from baseline score; Week 124: number analyzed (Participants) | 4
  Change from baseline score; Week 124 | -0.8 (1.26)

28. Secondary Outcome: Effect of SPN-812 on "Disruptions in Sleep Quality" (SDQ-4) Subscale in Adults With ADHD as Measured by the Symptoms of Depression Questionnaire (SDQ)
Description: An additional secondary endpoint was the change from baseline in the Symptoms of Depression Questionnaire (SDQ) "Disruptions in Sleep Quality" (SDQ-4) Subscale Score by visit. The SDQ is a 44-item self-rating scale assessing overall depression and 5 related symptoms/subscales, including 3 items related to disruptions in sleep quality (SDQ-4). Each item is rated on a 6-point scale based on a subject's perception in past month of what is normal (score = 2), what is better than normal (score = 1), and what is worse than normal (scores = 3-6). The sum of these 3 items yields the raw SDQ-4 subscale score (range: 3-18); a higher SDQ-4 subscale score indicates worse disruptions in sleep quality. Post-baseline raw SDQ-4 subscale scores are converted to a change from baseline score. A lower change from baseline SDQ-4 subscale score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
units on a scale
  Raw score; Baseline: number analyzed (Participants) | 158
  Raw score; Baseline | 7.9 (2.38)
  Change from baseline score; Week 2: number analyzed (Participants) | 14
  Change from baseline score; Week 2 | 1.1 (3.75)
  Change from baseline score; Week 4: number analyzed (Participants) | 121
  Change from baseline score; Week 4 | 0.1 (2.93)
  Change from baseline score; Week 12: number analyzed (Participants) | 109
  Change from baseline score; Week 12 | 0.1 (3.14)
  Change from baseline score; Week 20: number analyzed (Participants) | 95
  Change from baseline score; Week 20 | -0.2 (2.45)
  Change from baseline score; Week 28: number analyzed (Participants) | 79
  Change from baseline score; Week 28 | 0.0 (2.15)
  Change from baseline score; Week 36: number analyzed (Participants) | 67
  Change from baseline score; Week 36 | -0.3 (2.20)
  Change from baseline score; Week 44: number analyzed (Participants) | 59
  Change from baseline score; Week 44 | -0.6 (2.42)
  Change from baseline score; Week 52: number analyzed (Participants) | 51
  Change from baseline score; Week 52 | -0.6 (2.97)
  Change from baseline score; Week 60: number analyzed (Participants) | 39
  Change from baseline score; Week 60 | -0.5 (3.02)
  Change from baseline score; Week 68: number analyzed (Participants) | 35
  Change from baseline score; Week 68 | -1.2 (2.68)
  Change from baseline score; Week 76: number analyzed (Participants) | 33
  Change from baseline score; Week 76 | -0.7 (2.61)
  Change from baseline score; Week 84: number analyzed (Participants) | 29
  Change from baseline score; Week 84 | -1.6 (2.21)
  Change from baseline score; Week 92: number analyzed (Participants) | 25
  Change from baseline score; Week 92 | -1.4 (2.86)
  Change from baseline score; Week 100: number analyzed (Participants) | 13
  Change from baseline score; Week 100 | -0.2 (3.08)
  Change from baseline score; Week 108: number analyzed (Participants) | 9
  Change from baseline score; Week 108 | -1.0 (3.54)
  Change from baseline score; Week 116: number analyzed (Participants) | 7
  Change from baseline score; Week 116 | -0.9 (4.38)
  Change from baseline score; Week 124: number analyzed (Participants) | 4
  Change from baseline score; Week 124 | -1.8 (2.75)

29. Secondary Outcome: Effect of SPN-812 on "Appetite and Weight" (SDQ-5) Subscale in Adults With ADHD as Measured by the Symptoms of Depression Questionnaire (SDQ)
Description: An additional secondary endpoint was the change from baseline in the Symptoms of Depression Questionnaire (SDQ) "Appetite and Weight" (SDQ-5) Subscale Score by visit. The SDQ is a 44-item self-rating scale assessing overall depression and 5 related symptoms/subscales, including 4 items related to changes in appetite and weight (SDQ-5). Each item is rated on a 6-point scale based on a subject's perception in past month of what is normal (score = 2), what is better than normal (score = 1), and what is worse than normal (scores = 3-6). The sum of these 4 items yields the raw SDQ-5 subscale score (range: 4-24); a higher SDQ-5 subscale score indicates worse appetite and weight. Post-baseline raw SDQ-5 subscale scores are converted to a change from baseline score. A lower change from baseline SDQ-5 subscale score (<0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
units on a scale
  Raw score; Baseline: number analyzed (Participants) | 158
  Raw score; Baseline | 8.9 (1.32)
  Change from baseline score; Week 2: number analyzed (Participants) | 14
  Change from baseline score; Week 2 | 0.4 (0.93)
  Change from baseline score; Week 4: number analyzed (Participants) | 121
  Change from baseline score; Week 4 | 0.2 (1.47)
  Change from baseline score; Week 12: number analyzed (Participants) | 109
  Change from baseline score; Week 12 | 0.4 (1.48)
  Change from baseline score; Week 20: number analyzed (Participants) | 94
  Change from baseline score; Week 20 | 0.2 (1.51)
  Change from baseline score; Week 28: number analyzed (Participants) | 80
  Change from baseline score; Week 28 | 0.1 (1.62)
  Change from baseline score; Week 36: number analyzed (Participants) | 67
  Change from baseline score; Week 36 | 0.1 (1.89)
  Change from baseline score; Week 44: number analyzed (Participants) | 59
  Change from baseline score; Week 44 | 0.0 (1.40)
  Change from baseline score; Week 52: number analyzed (Participants) | 51
  Change from baseline score; Week 52 | 0.1 (1.55)
  Change from baseline score; Week 60: number analyzed (Participants) | 39
  Change from baseline score; Week 60 | 0.4 (1.39)
  Change from baseline score; Week 68: number analyzed (Participants) | 35
  Change from baseline score; Week 68 | 0.2 (1.57)
  Change from baseline score; Week 76: number analyzed (Participants) | 33
  Change from baseline score; Week 76 | 0.1 (1.20)
  Change from baseline score; Week 84: number analyzed (Participants) | 29
  Change from baseline score; Week 84 | 0.0 (1.09)
  Change from baseline score; Week 92: number analyzed (Participants) | 25
  Change from baseline score; Week 92 | 0.2 (1.46)
  Change from baseline score; Week 100: number analyzed (Participants) | 13
  Change from baseline score; Week 100 | -0.5 (0.78)
  Change from baseline score; Week 108: number analyzed (Participants) | 9
  Change from baseline score; Week 108 | -0.2 (1.39)
  Change from baseline score; Week 116: number analyzed (Participants) | 7
  Change from baseline score; Week 116 | -0.3 (1.50)
  Change from baseline score; Week 124: number analyzed (Participants) | 4
  Change from baseline score; Week 124 | 0.3 (1.26)

30. Secondary Outcome: Effect of SPN-812 on Overall Quality of Life in Adults With ADHD as Measured by the Adult ADHD Quality of Life Scale (AAQoL)
Description: An additional secondary endpoint was the change from baseline in the Adult ADHD Quality of Life Scale (AAQoL) Total score by visit. The AAQoL is a 29-item self-rating scale assessing how ADHD has impacted his/her quality of life. It includes 4 related aspects (subscales) of quality of life, including Life Productivity (11 items), Psychological Health (6 items), Relationships (5 items), and Life Outlook (7 items). Each item is rated on a 5-point scale based on a subject's perception in past 2 weeks, where 1 = Not at all/Never, 2 = A little, 3 = Somewhat, 4 = A lot, and 5 = Extremely/Very often. Item scores are transformed to a 0 to 100-point scale (1=0; 2=5; 3=50; 4=75; 5=100). The sum of the transformed 29 items is divided by 29 to yield the raw Total score (range: 0-100); a higher raw Total score represents better quality of life. Post-baseline raw Total scores are converted to a change from baseline (CFB) Total score. A higher CFB Total score (>0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: Safety Population (N), defined as subjects who signed Informed Consent and took at least 1 dose of SPN-812. At each Visit/Week, data is summarized with descriptive statistics for the number of subjects analyzed (n; subjects with a valid AAQoL assessment at baseline [pre-dosing] and at the respective post-baseline [after first dose] Visit/Week). Due to attrition and/or missing data, the number of subjects analyzed at each Visit/Week may be less than and unequal to Safety Population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
units on a scale
  Raw score; Baseline: number analyzed (Participants) | 128
  Raw score; Baseline | 54.9 (14.96)
  Change from baseline score; Week 2: number analyzed (Participants) | 10
  Change from baseline score; Week 2 | 4.5 (10.08)
  Change from baseline score; Week 4: number analyzed (Participants) | 97
  Change from baseline score; Week 4 | 10.3 (14.66)
  Change from baseline score; Week 12: number analyzed (Participants) | 87
  Change from baseline score; Week 12 | 12.2 (17.18)
  Change from baseline score; Week 20: number analyzed (Participants) | 73
  Change from baseline score; Week 20 | 13.6 (18.89)
  Change from baseline score; Week 28: number analyzed (Participants) | 62
  Change from baseline score; Week 28 | 16.6 (17.76)
  Change from baseline score; Week 36: number analyzed (Participants) | 52
  Change from baseline score; Week 36 | 14.7 (17.91)
  Change from baseline score; Week 44: number analyzed (Participants) | 43
  Change from baseline score; Week 44 | 17.7 (15.76)
  Change from baseline score; Week 52: number analyzed (Participants) | 38
  Change from baseline score; Week 52 | 16.7 (17.08)
  Change from baseline score; Week 60: number analyzed (Participants) | 30
  Change from baseline score; Week 60 | 16.6 (16.96)
  Change from baseline score; Week 68: number analyzed (Participants) | 26
  Change from baseline score; Week 68 | 16.7 (18.09)
  Change from baseline score; Week 76: number analyzed (Participants) | 26
  Change from baseline score; Week 76 | 17.2 (14.68)
  Change from baseline score; Week 84: number analyzed (Participants) | 22
  Change from baseline score; Week 84 | 17.3 (14.83)
  Change from baseline score; Week 92: number analyzed (Participants) | 18
  Change from baseline score; Week 92 | 18.2 (17.11)
  Change from baseline score; Week 100: number analyzed (Participants) | 9
  Change from baseline score; Week 100 | 14.5 (14.47)
  Change from baseline score; Week 108: number analyzed (Participants) | 6
  Change from baseline score; Week 108 | 15.8 (17.28)
  Change from baseline score; Week 116: number analyzed (Participants) | 5
  Change from baseline score; Week 116 | 14.5 (16.14)
  Change from baseline score; Week 124: number analyzed (Participants) | 1
  Change from baseline score; Week 124 | 6.0 (0)

31. Secondary Outcome: Effects of SPN-812 on "Life Productivity" Aspect of Quality of Life in Adults With ADHD as Measured by the Adult ADHD Quality of Life Scale (AAQoL)
Description: An additional secondary endpoint was the change from baseline in the Adult ADHD Quality of Life Scale (AAQoL) "Life Productivity" subscale score by visit. The AAQoL is a 29-item self-rating scale assessing how ADHD has impacted his/her quality of life, which includes 11 items related to Life Productivity. Each item is rated on a 5-point scale based on a subject's perception in past 2 weeks, where 1 = Not at all/Never, 2 = A little, 3 = Somewhat, 4 = A lot, and 5 = Extremely/Very often. Item scores are transformed to a 0 to 100-point scale (1=0; 2=5; 3=50; 4=75; 5=100). The sum of the transformed 11 items is divided by 11 to yield the raw "Life Productivity" subscale score (range: 0-100); the higher the "Life Productivity" subscale score, the better Life Productivity. Post-baseline raw "Life Productivity" subscale scores are converted to a change from baseline score. A higher change from baseline "Life Productivity" subscale score (>0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
units on a scale
  Raw score; Baseline: number analyzed (Participants) | 157
  Raw score; Baseline | 45.6 (21.27)
  Change from baseline score; Week 2: number analyzed (Participants) | 14
  Change from baseline score; Week 2 | 13.6 (17.19)
  Change from baseline score; Week 4: number analyzed (Participants) | 120
  Change from baseline score; Week 4 | 18.0 (19.79)
  Change from baseline score; Week 12: number analyzed (Participants) | 108
  Change from baseline score; Week 12 | 18.9 (22.07)
  Change from baseline score; Week 20: number analyzed (Participants) | 94
  Change from baseline score; Week 20 | 21.3 (26.26)
  Change from baseline score; Week 28: number analyzed (Participants) | 80
  Change from baseline score; Week 28 | 24.4 (23.91)
  Change from baseline score; Week 36: number analyzed (Participants) | 67
  Change from baseline score; Week 36 | 23.5 (25.21)
  Change from baseline score; Week 44: number analyzed (Participants) | 59
  Change from baseline score; Week 44 | 24.1 (22.86)
  Change from baseline score; Week 52: number analyzed (Participants) | 51
  Change from baseline score; Week 52 | 25.8 (24.38)
  Change from baseline score; Week 60: number analyzed (Participants) | 39
  Change from baseline score; Week 60 | 26.9 (25.13)
  Change from baseline score; Week 68: number analyzed (Participants) | 36
  Change from baseline score; Week 68 | 26.5 (22.23)
  Change from baseline score; Week 76: number analyzed (Participants) | 33
  Change from baseline score; Week 76 | 26.2 (23.41)
  Change from baseline score; Week 84: number analyzed (Participants) | 29
  Change from baseline score; Week 84 | 27.2 (20.98)
  Change from baseline score; Week 92: number analyzed (Participants) | 24
  Change from baseline score; Week 92 | 26.5 (23.20)
  Change from baseline score; Week 100: number analyzed (Participants) | 13
  Change from baseline score; Week 100 | 25.5 (24.00)
  Change from baseline score; Week 108: number analyzed (Participants) | 9
  Change from baseline score; Week 108 | 32.1 (26.07)
  Change from baseline score; Week 116: number analyzed (Participants) | 7
  Change from baseline score; Week 116 | 30.2 (26.88)
  Change from baseline score; Week 124: number analyzed (Participants) | 3
  Change from baseline score; Week 124 | 39.4 (27.11)

32. Secondary Outcome: Effects of SPN-812 on "Psychological Health" Aspect of Quality of Life in Adults With ADHD as Measured by the Adult ADHD Quality of Life Scale (AAQoL)
Description: An additional secondary endpoint was the change from baseline in the Adult ADHD Quality of Life Scale (AAQoL) "Psychological Health" subscale score by visit. The AAQoL is a 29-item self-rating scale assessing how ADHD has impacted his/her quality of life, which includes 6 items related to Psychological Health. Each item is rated on a 5-point scale based on a subject's perception in past 2 weeks, where 1 = Not at all/Never, 2 = A little, 3 = Somewhat, 4 = A lot, and 5 = Extremely/Very often. Item scores are transformed to a 0 to 100-point scale (1=0; 2=5; 3=50; 4=75; 5=100). The sum of the transformed 6 items is divided by 6 to yield the raw "Psychological Health" subscale score (range: 0-100); the higher the subscale score, the better Psychological Health. Post-baseline raw "Psychological Health" subscale scores are converted to a change from baseline score. A higher change from baseline "Psychological Health" subscale score (>0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
units on a scale
  Raw score; Baseline: number analyzed (Participants) | 158
  Raw score; Baseline | 65.1 (19.54)
  Change from baseline score; Week 2: number analyzed (Participants) | 14
  Change from baseline score; Week 2 | 3.0 (15.63)
  Change from baseline score; Week 4: number analyzed (Participants) | 121
  Change from baseline score; Week 4 | 5.2 (18.45)
  Change from baseline score; Week 12: number analyzed (Participants) | 109
  Change from baseline score; Week 12 | 5.6 (21.38)
  Change from baseline score; Week 20: number analyzed (Participants) | 93
  Change from baseline score; Week 20 | 8.1 (17.97)
  Change from baseline score; Week 28: number analyzed (Participants) | 80
  Change from baseline score; Week 28 | 9.3 (20.49)
  Change from baseline score; Week 36: number analyzed (Participants) | 67
  Change from baseline score; Week 36 | 8.6 (18.47)
  Change from baseline score; Week 44: number analyzed (Participants) | 58
  Change from baseline score; Week 44 | 10.1 (19.17)
  Change from baseline score; Week 52: number analyzed (Participants) | 50
  Change from baseline score; Week 52 | 7.2 (19.47)
  Change from baseline score; Week 60: number analyzed (Participants) | 39
  Change from baseline score; Week 60 | 9.5 (17.78)
  Change from baseline score; Week 68: number analyzed (Participants) | 36
  Change from baseline score; Week 68 | 8.6 (20.51)
  Change from baseline score; Week 76: number analyzed (Participants) | 33
  Change from baseline score; Week 76 | 13.3 (18.29)
  Change from baseline score; Week 84: number analyzed (Participants) | 29
  Change from baseline score; Week 84 | 14.1 (16.72)
  Change from baseline score; Week 92: number analyzed (Participants) | 24
  Change from baseline score; Week 92 | 16.0 (18.33)
  Change from baseline score; Week 100: number analyzed (Participants) | 13
  Change from baseline score; Week 100 | 13.5 (17.36)
  Change from baseline score; Week 108: number analyzed (Participants) | 9
  Change from baseline score; Week 108 | 15.3 (22.92)
  Change from baseline score; Week 116: number analyzed (Participants) | 7
  Change from baseline score; Week 116 | 16.1 (17.42)
  Change from baseline score; Week 124: number analyzed (Participants) | 4
  Change from baseline score; Week 124 | 22.9 (21.11)

33. Secondary Outcome: Effects of SPN-812 on "Life Outlook" Aspect of Quality of Life in Adults With ADHD as Measured by the Adult ADHD Quality of Life Scale (AAQoL)
Description: An additional secondary endpoint was the change from baseline in the Adult ADHD Quality of Life Scale (AAQoL) "Life Outlook" subscale score by visit. The AAQoL is a 29-item self-rating scale assessing how ADHD has impacted his/her quality of life, which includes 7 items related to Life Outlook. Each item is rated on a 5-point scale based on a subject's perception in past 2 weeks, where 1 = Not at all/Never, 2 = A little, 3 = Somewhat, 4 = A lot, and 5 = Extremely/Very often. Item scores are transformed to a 0 to 100-point scale (1=0; 2=5; 3=50; 4=75; 5=100). The sum of the transformed 7 items is divided by 7 to yield the raw "Life Outlook" subscale score (range: 0-100); the higher the subscale score, the better Life Outlook. Post-baseline raw "Life Outlook" subscale scores are converted to a change from baseline score. A higher change from baseline "Life Outlook" subscale score (>0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
units on a scale
  Raw score; Baseline: number analyzed (Participants) | 129
  Raw score; Baseline | 56.0 (14.52)
  Change from baseline score; Week 2: number analyzed (Participants) | 11
  Change from baseline score; Week 2 | -3.9 (16.63)
  Change from baseline score; Week 4: number analyzed (Participants) | 98
  Change from baseline score; Week 4 | 3.1 (16.05)
  Change from baseline score; Week 12: number analyzed (Participants) | 88
  Change from baseline score; Week 12 | 6.7 (17.18)
  Change from baseline score; Week 20: number analyzed (Participants) | 75
  Change from baseline score; Week 20 | 7.0 (20.82)
  Change from baseline score; Week 28: number analyzed (Participants) | 63
  Change from baseline score; Week 28 | 8.8 (21.02)
  Change from baseline score; Week 36: number analyzed (Participants) | 52
  Change from baseline score; Week 36 | 5.6 (20.79)
  Change from baseline score; Week 44: number analyzed (Participants) | 44
  Change from baseline score; Week 44 | 10.1 (18.37)
  Change from baseline score; Week 52: number analyzed (Participants) | 38
  Change from baseline score; Week 52 | 8.6 (18.76)
  Change from baseline score; Week 60: number analyzed (Participants) | 30
  Change from baseline score; Week 60 | 9.6 (22.77)
  Change from baseline score; Week 68: number analyzed (Participants) | 26
  Change from baseline score; Week 68 | 12.2 (23.61)
  Change from baseline score; Week 76: number analyzed (Participants) | 26
  Change from baseline score; Week 76 | 11.8 (13.28)
  Change from baseline score; Week 84: number analyzed (Participants) | 22
  Change from baseline score; Week 84 | 9.1 (14.90)
  Change from baseline score; Week 92: number analyzed (Participants) | 18
  Change from baseline score; Week 92 | 10.3 (12.90)
  Change from baseline score; Week 100: number analyzed (Participants) | 9
  Change from baseline score; Week 100 | 14.3 (17.03)
  Change from baseline score; Week 108: number analyzed (Participants) | 6
  Change from baseline score; Week 108 | 9.5 (16.39)
  Change from baseline score; Week 116: number analyzed (Participants) | 5
  Change from baseline score; Week 116 | 7.1 (12.11)
  Change from baseline score; Week 124: number analyzed (Participants) | 2
  Change from baseline score; Week 124 | -1.8 (17.68)

34. Secondary Outcome: Effects of SPN-812 on "Relationships" Aspect of Quality of Life in Adults With ADHD as Measured by the Adult ADHD Quality of Life Scale (AAQoL)
Description: An additional secondary endpoint was the change from baseline in the Adult ADHD Quality of Life Scale (AAQoL) "Relationships" subscale score by visit. The AAQoL is a 29-item self-rating scale assessing how ADHD has impacted his/her quality of life, which includes 5 items related to Relationships. Each item is rated on a 5-point scale based on a subject's perception in past 2 weeks, where 1 = Not at all/Never, 2 = A little, 3 = Somewhat, 4 = A lot, and 5 = Extremely/Very often. Item scores are transformed to a 0 to 100-point scale (1=0; 2=5; 3=50; 4=75; 5=100). The sum of the transformed 5 items is divided by 5 to yield the raw "Relationships" subscale score (range: 0-100); the higher the subscale score, the better the Relationships. Post-baseline raw "Relationships" subscale scores are converted to a change from baseline score. A higher change from baseline "Relationships" subscale score (>0) represents a better outcome.
Time Frame: Baseline and Week 2, 4, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 108, 116, and 124
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 159
units on a scale
  Raw score; Baseline: number analyzed (Participants) | 157
  Raw score; Baseline | 64.7 (19.78)
  Change from baseline score; Week 2: number analyzed (Participants) | 13
  Change from baseline score; Week 2 | 6.9 (18.09)
  Change from baseline score; Week 4: number analyzed (Participants) | 120
  Change from baseline score; Week 4 | 6.7 (19.29)
  Change from baseline score; Week 12: number analyzed (Participants) | 108
  Change from baseline score; Week 12 | 7.2 (21.57)
  Change from baseline score; Week 20: number analyzed (Participants) | 94
  Change from baseline score; Week 20 | 10.8 (20.34)
  Change from baseline score; Week 28: number analyzed (Participants) | 78
  Change from baseline score; Week 28 | 10.7 (19.93)
  Change from baseline score; Week 36: number analyzed (Participants) | 66
  Change from baseline score; Week 36 | 10.1 (22.27)
  Change from baseline score; Week 44: number analyzed (Participants) | 57
  Change from baseline score; Week 44 | 10.7 (20.36)
  Change from baseline score; Week 52: number analyzed (Participants) | 50
  Change from baseline score; Week 52 | 13.3 (19.73)
  Change from baseline score; Week 60: number analyzed (Participants) | 38
  Change from baseline score; Week 60 | 11.8 (19.26)
  Change from baseline score; Week 68: number analyzed (Participants) | 35
  Change from baseline score; Week 68 | 11.9 (20.37)
  Change from baseline score; Week 76: number analyzed (Participants) | 32
  Change from baseline score; Week 76 | 14.4 (20.63)
  Change from baseline score; Week 84: number analyzed (Participants) | 28
  Change from baseline score; Week 84 | 12.7 (21.58)
  Change from baseline score; Week 92: number analyzed (Participants) | 24
  Change from baseline score; Week 92 | 11.7 (19.26)
  Change from baseline score; Week 100: number analyzed (Participants) | 12
  Change from baseline score; Week 100 | 13.8 (17.47)
  Change from baseline score; Week 108: number analyzed (Participants) | 8
  Change from baseline score; Week 108 | 11.9 (18.11)
  Change from baseline score; Week 116: number analyzed (Participants) | 7
  Change from baseline score; Week 116 | 5.7 (12.05)
  Change from baseline score; Week 124: number analyzed (Participants) | 4
  Change from baseline score; Week 124 | 18.8 (24.28)

ADVERSE EVENTS:
Time Frame: up to 156 weeks
Description: Number of subjects is based on Safety Population (defined as subjects who took at least one dose of SPN-812)
Arm/Group | Open-Label Treatment
All-Cause Mortality (participants affected / at risk) | 0/159
Serious Adverse Events (participants affected / at risk) | 2/159
Other Adverse Events (participants affected / at risk) | 114/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Treatment (N=159)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Treatment (N=159)
Insomnia (Psychiatric disorders) | 22 (26)
Nausea (Gastrointestinal disorders) | 22 (27)
Headache (Nervous system disorders) | 17 (23)
Fatigue (General disorders) | 16 (19)
Corona virus infection (Infections and infestations) | 11 (12)
Anxiety (Psychiatric disorders) | 10 (10)
Dry mouth (Gastrointestinal disorders) | 8 (9)
Vomiting (Gastrointestinal disorders) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT04143217/Prot_002.pdf
  • Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT04143217/SAP_003.pdf